Title: A proof-of-concept, randomized, double-blind, placebo-controlled, Phase

2a study to assess the prophylactic antiviral activity against influenza, safety, tolerability, and pharmacokinetics of CD388 via a human viral

challenge model

NCT Number: NCT05523089

**Document Date:** 25 JUL 2023



## **Statistical Analysis Plan**



# Cidara Therapeutics, Inc. CDT-CSP-001 / CD388.SQ.2.02

A proof-of-concept, Randomised, Double-blind, Placebo-controlled, Phase 2a Study to assess the prophylactic antiviral activity against influenza, safety, tolerability and pharmacokinetics of CD388 via a human viral challenge model

## **Statistical Analysis Plan**

Version: v2

Date: 25Jul2023

Antoinette Anger Venn Life Sciences Biometry Services 24-26 rue de la Pépinière | 75008 Paris | France Tel Office: +33 (0)1 40 21 04 10

antoinette.anger@vennlife.com
http://www.vennlifesciences.com

This document is to be considered CONFIDENTIAL and is for the sole use and review by Cidara Therapeutics, Inc. to whom the document is addressed. This document may not be shared with third parties, including but not limited to contract research organisations and other pharmaceutical service providers, without the express written permission of Venn Life Sciences.




# Statistical Analysis Plan

# Signatures and version history

## **Signature**

| Venn Life Sciences | | | |
|---|---|---|---|
| | Name Function Date and Signature | | |
| Written by | Antoinette<br>Anger | Associate Head of<br>Statistics | DocuSigned by: Intoinette Inger Signer Name: Antoinette Anger Signing Reason: I am the author of this document Signing Time: 25-Jul-2023 8:12:21 AM PDT D8AB006C654B4E9CB5F4CE85D0841495 |
| Reviewed<br>by | Elodie<br>Blondiaux | Methodology &<br>Biometrics<br>Consultant | DocuSigned by: Elodic Blondiaux Signer Name: Elodie Blondiaux Signing Reason: I have reviewed this document Signing Time: 25-Jul-2023 5:13:38 PM CEST 4832F141BED940A2A126AB01E747A040 |

| | Cidara | | |
|---|---|---|---|
| | Name | Function | Date and Signature |
| Approved by | Ozlem Equils | Medical Monitor | DocuSigned by: Signer Name: Ozlem Equils, MD Signing Reason: I approve this document Signing Time: 25-Jul-2023 8:08:25 AM PDT 8C319F80E19A475B89044981B91CEB55 |

## **Document version history**

| Version Date | | Author | Modifications since previous version |
|---|---|---|---|
| V1 | 16DEC2022 | Antoinette Anger | NA (initial release) |
| V2 | 25JUL2023 | Antoinette Anger | Update to section 12.3 |




# **Statistical Analysis Plan**

## **Table of Contents**

| Α | RRKEVIA | TIONS AND DEFINITIONS | 6 |
|---|---------|-----------------------------------------------------------|----|
| 1 | INTR | ODUCTION | 8 |
| 2 | HIGH | ILIGHTS FROM STUDY PROTOCOL | 8 |
| | 2.1 | BACKGROUND/RATIONALE | 8 |
| | 2.2 | STUDY OBJECTIVES AND ENDPOINTS | |
| | 2.2.1 | Primary objective and endpoint | 8 |
| | 2.2.2 | | |
| | 2.2.3 | | |
| | 2.3 | Investigational plan | 12 |
| | 2.3.1 | Study design and study assessments | 12 |
| | 2.3.2 | Randomization | 14 |
| | 2.3.3 | Determination of sample size | 16 |
| 3 | ANA | LYSIS DATASETS | 16 |
| | 3.1 | PROTOCOL DEVIATIONS | 16 |
| | 3.1.1 | Major protocol deviations | 16 |
| | 3.1.2 | | |
| | 3.2 | STUDY TREATMENT DISCONTINUATIONS - STUDY DISCONTINUATIONS | |
| | 3.2.1 | Participant Withdrawal | 17 |
| | 3.2.2 | Participant Discontinuation | 17 |
| | 3.2.3 | Lost to Follow up | 17 |
| | 3.2.4 | Participant Replacement Policy | 17 |
| | 3.3 | ANALYSIS SET DEFINITIONS | 17 |
| | 3.3.1 | Enrolled analysis set | 17 |
| | 3.3.2 | Intent-to-treat (ITT) analysis set | 17 |
| | 3.3.3 | Intent-to-treat Infected (ITT-I) analysis set | 17 |
| | 3.3.4 | Per-protocol (PP) analysis set | 18 |
| | 3.3.5 | Safety (SAF) analysis set | 18 |
| | 3.3.6 | Pharmacokinetic (PK) analysis set | 18 |
| 4 | ENDI | POINTS FOR ANALYSIS | 18 |
| | 4.1 | EFFICACY ENDPOINTS | 18 |
| | 4.1.1 | Primary efficacy endpoint | 18 |
| | 4.1.2 | Secondary efficacy endpoints | 18 |
| | 4.1.3 | Tertiary/Exploratory efficacy endpoints | 21 |
| | 4.2 | SAFETY ENDPOINTS | 23 |
| | 4.2.1 | Adverse events | 23 |
| | 4.2.2 | Laboratory endpoints | 24 |
| | 4.2.3 | Other safety endpoints | 24 |
| | 4.2.4 | Concomitant medications | 26 |
| 5 | STAT | ISTICAL AND ANALYTICAL METHODS | 27 |
| | 5.1 | GENERAL CONSIDERATIONS | 27 |



# **Statistical Analysis Plan**

| | 5.1.1 | Presentation of results | 27 |
|---|---|---|---|
| | 5.1.2 | Significance testing and estimation | 27 |
| | 5.2 | SEQUENCE OF ANALYSES | 28 |
| | 5.3 | PLANNED ANALYSIS | 28 |
| | 5.3.1 | Participant disposition and study discontinuations | 28 |
| | 5.3.2 | Protocol deviations | 28 |
| | 5.3.3 | Demographics and baseline characteristics | 29 |
| | 5.3.4 | Medical history – Prior medications | 29 |
| | 5.3.5 | Concomitant medications | 29 |
| | 5.3.6 | Spirometry | 30 |
| | 5.3.7 | Efficacy analyses | 30 |
| | 5.3.8 | Safety analyses | 36 |
| 6 | DATA | A HANDLING CONVENTIONS | 42 |
| | 6.1 | DEFINITIONS | 42 |
| | 6.1.1 | | |
| | 6.1.2 | - | |
| | 6.2 | RETEST, OUTLIERS | 43 |
| | 6.2.1 | Retests | 43 |
| | 6.2.2 | Outliers | 43 |
| | 6.3 | VISIT WINDOWS, UNSCHEDULED VISITS | 43 |
| | 6.3.1 | Windows for time points | 43 |
| | 6.3.2 | Unscheduled visits | 43 |
| | 6.4 | MISSING DATA AND ANALYSIS RULES | 43 |
| | 6.4.1 | Missing data | 43 |
| | 6.4.2 | Analysis rules | 44 |
| 7 | DERI | VED DATA | 45 |
| 8 | INTE | RIM ANALYSIS | 46 |
| 9 | <b>STΔT</b> | ISTICAL/ANALYTICAL ISSUES | 47 |
| | | ADJUSTMENTS FOR COVARIATES | |
| | _ | HANDLING OF DROPOUTS OR MISSING DATA | |
| | | Interim Analyses and Data Monitoring | |
| | | MULTICENTRE STUDIES | |
| | | MULTIPLE COMPARISON/MULTIPLICITY | |
| | | Use of an "Efficacy Subset" of Participants | |
| | | ACTIVE-CONTROL STUDIES INTENDED TO SHOW EQUIVALENCE | |
| | | EXAMINATION OF SUBGROUPS | |
| | | IFICATIONS FROM THE STATISTICAL SECTION OF THE PROTOCOL | |
| 10 | | | |
| 11 | | WARE DOCUMENTATION | |
| 12 | TABL | ES, FIGURES AND LISTINGS | 49 |
| | 12.1 | LIST OF TABLES | 49 |
| | 12.2 | LIST OF FIGURES | 49 |





# **Statistical Analysis Plan**

| 1 | 2.3 | LIST OF LISTINGS | .49 |
|----|------|------------------|-----|
| 13 | REFE | ERENCES | 50 |
| 14 | SCHI | EDULE OF EVENTS | 51 |



Venn Life Sciences Think Research

Document Version: v2

## **Statistical Analysis Plan**

#### Abbreviations and definitions

ADA Anti-drug antibody ΑE Adverse Event

ALT Alanine aminotransferase **AST** Aspartate aminotransferase

aPTT **Activated Partial Thromboplastin Time** ATC **Anatomical Therapeutic Chemical** 

AUC Area Under the Curve **BDRM** Blind Data Review Meeting

**BHCG** Beta-Human chorionic gonadotropin

BMI **Body Mass Index** BP **Blood Pressure** Bpm Beats per minute CI Confidence interval CM **Concomitant Medication** 

CRO **Contract Research Organization** 

CS **Clinically Significant** 

**CTCAE** Common Terminology Criteria for Adverse Events

**DAIDS** Division of AIDS **ECG** Electrocardiogram **EOS End of Study** 

FEV1 Forced expiratory volume (in 1 second)

**FSH** Follicle-stimulating hormone

FVC Forced vital capacity

Gamma-Glutamyl Transferase **GGT** HIV Human immunodeficiency virus

HR **Heart Rate** 

**HVC Human Viral Challenge** 

**ICH** International Council of Harmonization

**IMP Investigational Medical Product** 

ΙP **Investigational Product** ITT Intention-to-Treat

ITT-I Intention-to-Treat infected LDH Lactate Dehydrogenase LLN **Lower Limit Normal** LLOD Lower limit of detection LLOQ Lower limit of quantification LRT **Lower Respiratory Tract** 

MedDRA Medical Dictionary for Regulatory Activities

МН **Medical History** Ms Millisecond

NCS Non-Clinically Significant Ы **Principal Investigator** PK Pharmacokinetic(s)

PP Per-Protocol




## CIDARA\_CDT-CSP-001\_SAP\_V2\_Final\_25Jul23


## **Statistical Analysis Plan**

PT Prothrombine Time
PT Preferred Term

Q1 First quartile – 25th percentile
Q3 Third quartile – 75th percentile

RR Respiratory Rate

qRT PCR quantitative Reverse Transcriptase-Polymerase Chain Reaction

SAE Serious Adverse Event

SAF Safety dataset

SAP Statistical Analysis Plan
SD Standard Deviation
SOC System Organ Class

SOP Standard operating procedure

SoE Schedule of events
TBD To be defined

TEAE Treatment-Emergent Adverse Event

TESAE Treatment-Emergent Serious Adverse Event

TFL Tables Figures Listings
TSS Total Symptom Score
ULN Upper Limit Normal
URT Upper Respiratory Tract

VL Viral load

WHO Word Health Organization




## **Statistical Analysis Plan**

#### 1 Introduction

This document is the statistical analysis plan (SAP) for the CDT-CSP-001 study. The purpose of this SAP, developed following the International Council of Harmonization (ICH) E9 guideline, is to provide a comprehensive and detailed description of the statistical analyses that will be carried out to assess the clinical efficacy and safety of the study treatment, as outlined in the study protocol version 1.0, dated June 7, 2022. The SAP pre-specifies the statistical approaches to be used and is validated prior to the first interim analysis and the unblinding of the randomisation schedule, to ensure the credibility of the study findings.

## 2 Highlights from study protocol

## 2.1 Background/Rationale

Full details on the background and rationale for the study are provided in Sections 2.1 to 2.3 of the protocol.

The purpose of this Phase 2a study is to evaluate the safety, tolerability, and prophylactic antiviral efficacy of CD388 compared to placebo in healthy adult participants who have not received an influenza vaccine and who are naïve to the influenza H3N2 A/Perth/16/2009 challenge virus as defined by HA titres ≤1:10.

## 2.2 Study Objectives and Endpoints

## 2.2.1 Primary objective and endpoint

To evaluate the prophylactic antiviral effect of CD388 compared to placebo when treatment is initiated prior to administration with the influenza H3N2 A/Perth/16/2009 challenge virus by assessing the reduction of area under the viral load-time curve (VLAUC) measured by quantitative reverse transcriptase-polymerase chain reaction (qRT PCR) on nasal samples starting a day post viral challenge (Day 1, pm) up to Day 8 (am) in treated participants vs. placebo participants.

## 2.2.2 Secondary objectives and endpoints

## 2.2.2.1 Efficacy

To evaluate the antiviral effect of CD388 in:

- reducing or shortening viral shedding after influenza viral challenge compared to placebo by assessing the following endpoints
  - Peak viral load of influenza as defined by the maximum viral load determined by quantifiable qRT-PCR measurements in nasal samples from Day 1 (pm) up to Day 8 (am).
  - Time (hours) to confirmed negative test by quantifiable qRT-PCR measurements in nasal samples from Day 1 (pm) to first confirmed undetectable assessment after peak measure.


## **Statistical Analysis Plan**

- reducing or shortening culturable/replicating virus after influenza viral challenge compared to placebo by assessing the following endpoints:
  - VL-AUC of influenza challenge virus as determined by viral culture on nasal samples, from Day 1 (pm) up to Day 8 (am).
  - Peak viral load of influenza as defined by the maximum viral load determined by quantitative viral culture measurements in nasal samples from Day 1 (pm) up to Day 8 (am).
  - Time (hours) to confirmed negative test by quantifiable viral culture measurements in nasal samples from Day 1 (pm) to first confirmed undetectable assessment after peak measure.
- reducing clinical symptoms due to influenza viral challenge compared to placebo by assessing the following endpoints:
  - Area under the curve over time of total clinical symptoms score (TSS-AUC) as measured by graded symptom scoring system collected 3 times daily from Day 1 (am) up to Day 8 (am).
  - Peak symptoms diary card score: peak of total clinical symptoms (TSS) as measured by graded symptom scoring system collected 3 times daily from Day 1 (am) up to Day 8 (am).
  - Peak daily symptom score: individual maximum daily sum of symptom score from Day 1 up to Day 8.
  - Time to symptom resolution as measured by graded daily symptom score system from time of peak daily symptom score to time of returning to baseline score.
- reducing the incidence of influenza infection due to influenza viral challenge, compared to placebo by assessing the following endpoints:
  - RT-PCR-confirmed influenza infection, defined as 2 quantifiable (≥ lower limit of quantification [LLOQ]) qRT-PCR measurements (reported on 2 or more independent samples over 2 days), from Day 1 (pm) up to Day 8 (am).
  - Occurrence of at least 1 positive quantitative (≥LLOQ) cell culture measurement in nasal samples, from Day 1 (pm) up to Day 8 (am).
  - RT-PCR-confirmed symptomatic influenza infection, defined as:
    - RT-PCR-confirmed influenza infection (2 quantifiable [≥LLOQ] qRT-PCR measurements [reported on 2 or more independent samples over 2 days]), from Day 1 (pm) up to Day 8 (am), AND
    - Symptoms ≥2 at a single time point (from Day 1 to Day 8)
  - RT-PCR-confirmed moderately severe symptomatic influenza infection, defined as:
    - RT-PCR-confirmed influenza infection (2 quantifiable [≥LLOQ] qRT-PCR measurements [reported on 2 or more independent samples over 2 days]), from Day 1 (pm) up to Day 8 (am), AND


- Any symptoms of grade  $\geq 2$  at a single time point (from Day 1 to Day 8).
- Culture lab-confirmed symptomatic influenza infection, defined as:
  - Lab-confirmed culturable influenza infection (1 quantifiable [≥LLOQ] cell culture measurement), from Day 1 (pm) up to Day 8 (am), AND
  - Symptoms ≥2 at a single time point (from Day 1 to Day 8).

## 2.2.2.2 Safety

To evaluate the safety of CD388 when compared to placebo on the basis of the following endpoints:

- Occurrence of solicited Adverse Events (AEs) from subcutaneous dosing up to Day 0.
- Occurrence of unsolicited AEs from subcutaneous dosing up to Day 28 (±3 days).
- Occurrence of unsolicited AEs from subcutaneous dosing up to the final follow-up visit (Day 180 ±14 days).

## 2.2.3 Tertiary/exploratory objectives\*

To further evaluate the antiviral effect of CD388 in:

- reducing or shortening viral shedding after influenza viral challenge compared to placebo by assessing the following endpoint:
  - Duration of quantifiable influenza qRT-PCR measurements in nasal samples from Day 1 (pm) up to Day 8 (am). Duration is defined as the time (hours) from first detectable until first confirmed undetectable assessment after their peak measure (after which no further virus is detected).
- reducing or shortening culturable/replicating virus after influenza viral challenge compared to placebo by assessing the following endpoint:
  - Duration of quantitative influenza viral culture measurements in nasal samples from Day 1 (pm) up to Day 8 (am). Duration is defined as the time (hours) from first detectable until first confirmed undetectable assessment after their peak measure (after which no further virus is detected).
- reducing clinical symptoms due to influenza viral challenge compared to placebo by assessing by assessing the following endpoints:
  - Time to peak as measured by graded daily symptom score system (from Day 1 [am] to the time of peak daily symptom score).
  - Number (%) of participants with symptom scored grade 2 or higher, from Day 1 (am) up to Day 8 (am).
  - Number (%) of participants with symptom scored grade 2 or higher by time point, from Day 1 (am) up to Day 8 (am).
- reducing the incidence of influenza infection due to influenza viral challenge, compared to placebo by assessing by assessing the following endpoints:
  - Number (%) of participants with lab-confirmed infection and fever (≥37.9°C).


## **Statistical Analysis Plan**

- Further sensitivity analysis may be performed on the above qRT-PCR-related incidence endpoints where detection by qRT-PCR is reported above the lower limit of detection (LLOD) instead of the LLOQ.
- reducing nasal discharge compared to placebo by assessing the following endpoints:
  - o Total weight of mucus produced from Day 1 (am) up to Day 8 (am).
  - Total number of facial tissues used by participants from Day 1 (am) up to Day 8 (am).
- reducing incidence of community-acquired influenza infection compared to placebo by assessing the following endpoint:
  - Laboratory--confirmed symptomatic influenza infection (community acquired), defined as:
    - Self-reported influenza-like symptoms, AND
    - Community acquired (not challenge virus) laboratory-confirmed influenza infection PCR measurement and/or lateral flow positive, or other equivalent) reported on any occasion from discharge from quarantine up to Day 90 and/or up to Day 180 (±14 days).
- To monitor the safety of the challenge virus in the basis of the the following endpoint:
  - o Occurrence of unsolicited AEs from virus challenge (Day 0) up to Day 28.
- To evaluate the plasma PK of CD388 based on the following endpoints:
  - O Pharmacokinetic (PK) parameters following CD388 administration will be determined as appropriate from the available data including: maximum plasma concentration (Cmax), time to maximum plasma concentration (Tmax), area under the plasma concentration-time curve from time 0 to time of last quantifiable sample (AUCO-t), and area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUCO-∞).
- To explore CD388 concentrations in nasopharyngeal swab samples
- To explore PK/PD of CD388:
  - Plasma concentration at specific time points, or PK parameters across dose arms, will be compared to viral or symptomatic endpoints in an effort to characterise the exposure response of CD388, and will be reported separately
- To explore cytokines and chemokines in nasal samples:
  - Cytokine/chemokine levels may be explored in nasal samples, related to CD388 and infection.


- To explore cytokines and chemokines in serum samples:
  - Cytokine/chemokine levels may be explored in serum samples, related to CD388 and infection
- To explore markers associated with the effect of CD388 or with infection:
  - Gene expression (messenger RNA [mRNA]) in whole blood
- To explore viral resistance markers in influenza viral positive nasal samples:
  - Viral resistance markers relevant for CD388.

## 2.3 Investigational plan

## 2.3.1 Study design and study assessments

This is a single-centre, randomised, double-blind, placebo-controlled, proof-of-concept study in healthy adult male and female participants 18 to 55 years of age, inclusive, utilising:

- IMP (active): a single subcutaneous dose of CD388 liquid for injection
- IMP (placebo): a single subcutaneous dose of sterile normal saline for injection
- Challenge agent: influenza H3N2 A/Perth/16/2009 challenge strain, ~10<sup>5.5</sup> tissue culture infective dose (50%) (TCID<sub>50</sub>), intranasally administered

The primary goal of this Phase 2a study is to assess the prophylactic antiviral activity against influenza, safety, tolerability, and PK of CD388 via a HVC model, and to explore the impact of dose levels on efficacy. Each participant will receive a single administration of CD388 or placebo; multiple dose levels of CD388 may be evaluated.

Participants will be recruited based upon the following criteria: Healthy adult male and female participants aged between 18 to 55 years, inclusive, with a total body weight  $\geq$ 50 kg and body mass index (BMI)  $\geq$ 18 kg/m2 and  $\leq$ 35kg/m2, who have been determined to be sero-suitable with regard to pre-existing antibody levels to the influenza H3N2 A/Perth/16/2009 challenge virus.

A total of up to 168 participants is planned to be enrolled in this study in up to 2 cohorts. Cohort 1 will consist of up to 90 participants that will be enrolled simultaneously; a placebo arm (Arm 1, n= up to 30) and two CD388 dose arms (Arm 2 [150 mg CD388, n= up to 30] and Arm 3 [50 mg CD388, n= up to 30]). Cohort 2 details will be confirmed further to interim analysis as described below. Cohort 2 may include extension of the arms in Cohort 1 or include additional dose levels not exceeding 150 mg.

Participants will receive CD388 or placebo prior to being inoculated with the influenza challenge virus and will undergo assessments as per Scheduled of Event (SoE). The timing of


<sup>\*</sup>Note that tertiary objectives and endpoints are optional and might be assessed only if needed; therefore, not all testing might be performed and reported.



## Statistical Analysis Plan

administration of CD388 or placebo is chosen so as to approximate Tmax of CD388 in plasma at the time of challenge virus inoculation.



- <sup>b</sup> Maximum dose will not exceed 150 mg. Doses may be adjusted based on PK results from Study CD388.IM.SQ.1.01
- <sup>c</sup> Analysis of participants from Cohort 1 informs on Cohort 2 in regards:
  - · dose levels to be investigated
  - N numbers per arm

## Figure 1: Overview of Study Design

The expected duration of study participation for a participant is approximately 9 months, with the following sequence and duration of study phases:

- Screening Phase: from Day -96 to Day -7/-6 quarantine admission. Historical generic screening data collected through the hVIVO generic screening process may be transferred to this study after the study-specific consent form has been signed by the participant.
- Inpatient Phase: Participants will be resident in the quarantine unit for approximately 16 days (from Day -7/-6 to Day 8). Procedures will include:

#### Pre-HVC:

- Admission to quarantine unit on Day -7/-6.
- Baseline assessments and randomisation will be conducted as per SoE up to Day -5, pre-dose.
- Administration of CD388 or placebo on Day -5.

#### HVC:

Influenza virus inoculation on Day 0.

## Post-HVC:

Day 1 onwards and each day – study assessments will be conducted as per SoE.




• Participants will be discharged from the quarantine unit on Day 8 (or may remain longer at the principal investigator's [PI's] discretion).

## - Outpatient Phase:

- Follow-up visit(s): Day 17 (±1 day), Day 28 (±3 days), Day 60 (±7 days), and Day 120 (±14 days).
- Final visit: Day 180 (±14 days).

## 2.3.1.1 Study Schematic: On-study Participant Progression



## NOTES:

#### 2.3.2 Randomization

In Cohort 1, the randomisation number encodes the participant's assignment to 1 of 3 study arms: placebo (Arm 1, n= 24 to 30), and two CD388 dose arms (150 mg CD388 [Arm 2, n=30]


<sup>\*</sup>Screening assessments (including repeats, as required), may be performed up to Day -7/-6, (quarantine admission) at the discretion of the PI/investigator and in accordance with the design of the study.

<sup>\*\*</sup>Release from quarantine is foreseen at Day 8 (8 days post inoculation) provided that, where appropriate, no virus is detected by qualitative virus antigen test (negative virus antigen test) and the participant has no clinically significant symptoms. If the participant continues to have clinically significant symptoms and/or detectable virus on Day 8, additional extended quarantine stay may be required at the discretion of the Pl/investigator.



## **Statistical Analysis Plan**

and 50 mg CD388, [Arm 3, n= 18 to 30]). This initial randomisation schedule, in use prior to Non-Substantial Amendment 03, used 2 varying block sizes (12 and 3) and 2 sets of randomisation ratios (4:5:3 and 1:0:2) to facilitate achieving the targeted sample sizes for the interim analysis.

| Block | | | | | Cumulative | | | |
|---|---|---|---|---|---|---|---|---|
| Block | Arm 1<br>Placebo | Arm 2<br>High dose<br>(150 mg CD388) | Arm 3<br>Low dose<br>(50 mg CD388) | Block size | Arm 1<br>Placebo | Arm 2<br>High dose<br>(150 mg CD388) | Arm 3<br>Low dose<br>(50 mg CD388) | Randomised |
| 1 | 4 | 5 | 3 | 12 | 4 | 5 | 3 | 12 |
| 2 | 4 | 5 | 3 | 12 | 8 | 10 | 6 | 24 |
| 3 | 4 | 5 | 3 | 12 | 12 | 15 | 9 | 36 |
| 4 | 4 | 5 | 3 | 12 | 16 | 20 | 12 | 48 |
| 5 | 4 | 5 | 3 | 12 | 20 | 25 | 15 | 60 |
| 6 | 4 | 5 | 3 | 12 | 24 | 30 | 18 | 72 |
| 7 | 1 | 0 | 2 | 3 | 25 | 30 | 20 | 75 |
| 8 | 1 | 0 | 2 | 3 | 26 | 30 | 22 | 78 |
| 9 | 1 | 0 | 2 | 3 | 27 | 30 | 24 | 81 |
| 10 | 1 | 0 | 2 | 3 | 28 | 30 | 26 | 84 |
| 22 | 1 | 0 | 2 | 3 | 29 | 30 | 28 | 87 |
| 23 | 1 | 0 | 2 | 3 | 30 | 30 | 30 | 90 |

At the time of Non-Substantial Amendment 03, this randomisation schedule was modified to ensure achievement of the largest possible sample-sizes in arm 1 (Placebo) and arm 2 (High dose) at the time of the planned first interim analysis. Participants enrolled under Non-Substantial Amendment 03 will be randomised 1:1 to either arm 1 (Placebo) or arm 2 (150 mg CD388) until Cohort 1 enrolment is complete. Afterwards, a new randomisation schedule will be prepared, taking into account the decisions taken based on the results of the first interim analysis.

Randomisation numbers will be assigned sequentially in ascending order; and once assigned, that randomisation number shall not be reassigned. The study site will keep a log of the randomisation number assigned to each participant.

A designated unblinded statistician, separate from the conduct or analysis of the study, will be responsible for the computer-generated randomisation schedule. Sealed copies of the randomisation code will be stored in a secure location.

Participants may be replaced in this study: If a participant discontinues from study intervention OR withdraws from the study for reasons not related to AEs, a replacement participant may be enrolled if deemed appropriate by the PI and sponsor.

If participants are replaced, the replacement participant will be assigned a new, unique randomisation number equalling the randomisation number of the replaced participant, plus




1000. This will ensure that the replacement participant receives the same allocated, blinded treatment as the participant who is being replaced.

#### 2.3.3 Determination of sample size

A total sample size of 168 participants is estimated to be sufficient to achieve the objectives of this study.

Depending on recruitment, the number enrolled at the planned first interim analysis is expected to be up to 30 participants in Arm 1 (placebo), Arm 2 (150 mg CD388), and Arm 3 (50 mg CD388). An example of sample size estimates for the interim analysis is shown below:

- The sample size of 30 participants per arm will have 95% power to detect a statistically significant difference between groups, using a Wilcoxon rank-sum test with a one-sided type-1 error rate of 0.025, assuming that the probability that the VL-AUC for a participant in Arm 2 (150 mg CD388) is less than the VL-AUC for a participant in Arm 1 (placebo) is 0.75.
- The sample size calculations used the method proposed in Shieh et al, 2009.

| Probability (AUC <sub>CD388</sub> < AUC <sub>Placebo</sub> ) | 0.60 | 0.65 | 0.70 | 0.75 | 0.80 |
|---|---|---|---|---|---|
| Power at Interim analysis | | | | | |
| Interim analysis Arm 1 n=30 vs Arm 2 n=30 | 0.259 | 0.515 | 0.785 | 0.951 | 0.996 |

AUC: area under the curve

## 3 Analysis datasets

## 3.1 Protocol deviations

All deviations will be determined to be major or minor according to the Project Management Plan. The impact of the deviation on the primary endpoint will be reviewed, during a blinded data review meeting before database lock and code break. Reasons for exclusion of participants from analysis sets due to major protocol deviations will be documented in the meeting minutes. A blinded data review meeting will be performed before each (interim) analysis.

## 3.1.1 Major protocol deviations

Major protocol deviations are defined as deviations liable to either impact the rights, safety or well-being of the participant or prevent or bias the interpretation of the efficacy results of the study. The following deviations may be considered as major (this list is not exhaustive)):

- Non-compliance with the inclusion or non-inclusion criteria
- Non-compliance with the randomisation procedure
- Non-compliance with study treatment
- Non-compliance with protocol-specified challenge virus inoculation procedures


- Missing data for the primary efficacy endpoint (or data collected for the primary efficacy endpoint in a manner diverging from protocol specifications)
- Intake of forbidden medication

#### 3.1.2 Minor protocol deviations

All deviations not identified as 'major' will be considered to be minor.

## 3.2 Study treatment discontinuations - Study discontinuations

## 3.2.1 Participant Withdrawal

See section 7.1 in the study Protocol.

#### 3.2.2 Participant Discontinuation

See section 7.2 in the study Protocol.

#### 3.2.3 Lost to Follow up

See section 7.3 in the study Protocol.

## 3.2.4 Participant Replacement Policy

See section 7.4 in the study Protocol.

#### 3.3 Analysis set definitions

Membership of participants in the per-protocol analysis set will be determined at planned blinded data review meetings, prior to any analysis. All other analysis sets will be determined programmatically based on data in the eCRF.

The primary efficacy analysis will be on the PP analysis set. The ITT analysis set will be used for supportive analyses on part of the primary and secondary efficacy endpoints. The safety evaluation will be performed on the safety analysis set.

## 3.3.1 Enrolled analysis set

All participants who sign the study-specific ICF.

#### 3.3.2 Intent-to-treat (ITT) analysis set

All participants randomly assigned and given study intervention. They will be analysed according to the treatment actually received

#### 3.3.3 Intent-to-treat Infected (ITT-I) analysis set

All participants randomly assigned and given the study intervention and infected with challenge agent as per the definition of laboratory-confirmed infection for this protocol, i.e., qRT-PCR-confirmed influenza infection, defined as 2 quantifiable (≥LLOQ) qRT-PCR measurements (2 quantifiable results reported within 4 consecutive scheduled assessments and from 2 independent samples), from Day 1 (pm) up to Day 8 (am).




## **Statistical Analysis Plan**

## 3.3.4 Per-protocol (PP) analysis set

All participants randomised, having received IMP (CD388/placebo), challenged with the study virus, who have a valid result for at least 80% of the planned qRT-PCR nasal samples from Day 1 (pm) up to Day 8 (am), i.e., at least 11 out of 14, and present no major deviations likely to impact the evaluation of the primary efficacy endpoint. All deviations and all cases who do not have at least 80% valid qRT-PCR result will be reviewed during blinded data review meetings (BDRM) and adjudicated as belonging to the PP set or not.

## 3.3.5 Safety (SAF) analysis set

All participants who received study intervention. Participants will be analysed according to the intervention they actually received.

#### 3.3.6 Pharmacokinetic (PK) analysis set

All participants randomly assigned to study intervention with at least 1 post-dose PK result.

## 4 Endpoints for analysis

The derivations of each endpoint for analysis are described in the following sections. In case of missing data, analysis rules are presented in Section 6.4.

## 4.1 Efficacy endpoints

## 4.1.1 Primary efficacy endpoint

The primary efficacy endpoint for the study is the total viral load AUC measured by qRT-PCR after viral challenge on Day 0: from (Day 1 pm) up to Day 8 (am).

The VL-AUC will be computed on the qRT PCR results from nasal samples collected twice daily starting with the first day post-viral challenge (Day 1 pm) up to discharge from quarantine (Day 8). The viral load data will be supplied as log10 copies/mL and the AUC will be calculated using the trapezium rule (method described in Section 7). The VL-AUC results will be expressed in log10 copies/mL \* day.

#### 4.1.2 Secondary efficacy endpoints

The secondary efficacy endpoints for the study are:

#### 4.1.2.1 Influenza infection

- Peak viral load of influenza as defined by the maximum viral load determined by quantifiable qRT-PCR measurements in nasal samples from Day 1 (pm) up to Day 8 (am) will be calculated per participant and will be supplied as log10 copies/mL.
- Time (hours) to confirmed negative test by quantifiable qRT-PCR measurements in nasal samples from Day 1 (pm) to first confirmed undetectable assessment (Result equal to Not detected, <LLOD) after peak measure (after which no further virus is detected). Participants who did not have a confirmed undetectable qRT-PCR assessment after their peak will be censored at their last detectable assessment. Participants who do not have a detectable qRT-PCR value during


## **Statistical Analysis Plan**

quarantine will be excluded from the analysis. In case of missing assessments, the LOCF type imputation will be used.

- VL-AUC of influenza challenge virus as determined by viral culture on nasal samples, from Day 1 (pm) up to Day 8 (am). The viral load data will be supplied as log10 PFU/mL and the AUC will be calculated using the trapezium rule (described in Section 7). The VL-AUC results will be expressed in log10 PFU/mL \* day.
- Peak viral load of influenza as defined by the maximum viral load determined by quantitative viral culture measurements in nasal samples from Day 1 (pm) up to Day 8 (am) will be calculated per participant and will be supplied as log10 PFU/mL.
- Time (hours) to confirmed negative test by quantifiable viral culture measurements in nasal samples from Day 1 (pm) to first confirmed undetectable assessment (Result equal to Not detected (<LLOD)) after peak measure. Participants who did not have a confirmed undetectable viral culture measurement after their peak will be censored at their last detectable assessment. Participants who do not have a detectable viral culture measure during quarantine will be excluded from the analysis. The number of these excluded participants will be displayed. In case of missing assessments, the LOCF type imputation will be used.</p>
- qRT-PCR-confirmed influenza infection, defined as 2 quantifiable (≥ lower limit of quantification [LLOQ]) qRT-PCR measurements (2 quantifiable results reported within 4 consecutive scheduled assessments and from 2 independent samples), from Day 1 (pm) up to Day 8 (am).

To define the condition 2 quantifiable results reported within 4 consecutive scheduled assessments and from 2 independent samples, we will use the following rule:

| Assessment 1 | Assessment 2 | Assessment 3 | Assessment 4 | Condition met? |
|---|---|---|---|---|
| Quantifiable | Quantifiable | Quantifiable | Quantifiable | Yes |
| Quantifiable | Not quantifiable | Quantifiable | Quantifiable | Yes |
| Quantifiable | Quantifiable | Not quantifiable | Quantifiable | Yes |
| Quantifiable | Quantifiable | Quantifiable | Not quantifiable | Yes |
| Quantifiable | Not quantifiable | Not quantifiable | Quantifiable | Yes |
| Quantifiable | Quantifiable | Not quantifiable | Not quantifiable | Yes |
| Quantifiable | Not quantifiable | Quantifiable | Not quantifiable | Yes |
| Quantifiable | Not quantifiable | Not quantifiable | Not quantifiable | No |
| Not quantifiable | Quantifiable | Quantifiable | Quantifiable | Yes |
| Not quantifiable | Not quantifiable | Quantifiable | Quantifiable | Yes |
| Not quantifiable | Quantifiable | Not quantifiable | Quantifiable | Yes |
| Not quantifiable | Quantifiable | Quantifiable | Not quantifiable | Yes |
| Not quantifiable | Not quantifiable | Not quantifiable | Quantifiable | No |
| Not quantifiable | Quantifiable | Not quantifiable | Not quantifiable | No |






## **Statistical Analysis Plan**

| Not quantifiable | Not quantifiable | Quantifiable | Not quantifiable | No |
|---|---|---|---|---|
| Not quantifiable | Not quantifiable | Not quantifiable | Not quantifiable | No |

In case of missing data, no imputation will be done.

- Occurrence of at least 1 positive quantitative (≥LLOQ) viral culture measurement in nasal samples, from Day 1 (pm) up to Day 8 (am).
- gRT-PCR-confirmed symptomatic influenza infection, defined as:
  - RT-PCR-confirmed influenza infection (2 quantifiable [≥LLOQ] qRT-PCR measurements [2 quantifiable results reported within 4 consecutive scheduled assessments and from 2 independent samples]), from Day 1 (pm) up to Day 8 (am) derived following the method above, AND
  - At least one TSS ≥2 at a single time point from Day 1 (pm) up to Day 8 (am)
- qRT-PCR-confirmed moderately severe symptomatic influenza infection, defined as:
  - RT-PCR-confirmed influenza infection (2 quantifiable [≥LLOQ] qRT-PCR measurements [2 quantifiable results reported within 4 consecutive scheduled assessments and from 2 independent samples]), from Day 1 (pm) up to Day 8 (am), AND
  - At least one single symptom of grade ≥2 at a single time point from Day 1 (pm) up to Day 8 (am)
- Culture lab-confirmed symptomatic influenza infection, defined as:
  - Lab-confirmed culturable influenza infection (1 quantifiable [≥LLOQ] cell culture measurement), from Day 1 (pm) up to Day 8 (am), AND
  - At least one total clinical symptom score (TSS) ≥2 at a single time point from Day 1 (pm) up to Day 8 (am)

## 4.1.2.2 Clinical Symptoms

- AUC over time of total clinical symptoms score (TSS-AUC) as measured by graded symptom scoring system collected 3 times daily from Day 1 (am) up to Day 8 (am).
   The method to derive the TSS is described in Section 7. The TSS-AUC will be calculated using the trapezium rule (method described also in Section 7)
- Peak symptoms diary card score: peak of TSS as measured by graded symptom scoring system collected 3 times daily from Day 1 (am) up to Day 8 (am). The TSS is calculated at each day and at each 3 timepoints. Per participant, the highest TSS will be determined between all calculated TSS from Day 1 (am) up to Day 8 (am).
- Peak daily symptom score: individual maximum daily sum of symptom score from Day 1 up to Day 8. The TSS is calculated at each day and at each 3 timepoints. Per participant and per day, the highest TSS will be selected between the 3 times daily.
- Time to symptom resolution as measured by graded daily symptom score system from time of peak daily symptom score to time of returning to baseline score is measured as the time (hours) from peak daily symptom score (as defined in the




## **Statistical Analysis Plan**

previous endpoint) until first time with TSS equal to the TSS at baseline after which no further increase above the baseline TSS is observed.

Participants who do not have a TSS equal to baseline TSS after their peak TSS will be censored at their last TSS. Participants who have the baseline TSS during the whole quarantine will be excluded from this analysis.

In case of missing TSS, we can consider several cases: If the missing values are not the last assessments, these missing values will be imputed by the previous not missing assessment. If the missing TSS values are the last measurements, the LOCF imputation method will be used. If the baseline score is missing, the baseline TSS will be imputed to 0.

## 4.1.3 Tertiary/Exploratory efficacy endpoints

 Duration of quantifiable influenza qRT-PCR measurements in nasal samples from Day 1 (pm) up to Day 8 (am). Duration is defined as the time (hours) from first quantifiable until first confirmed unquantifiable assessment after their peak measure (after which no further virus is detected).

In case of some unquantifiable assessment in-between series of one or more quantifiable assessments, the last quantifiable assessment of the last series is to be used as the end of the duration period. Participants who do not have a confirmed unquantifiable (i.e., <LLOQ, detected or not detected) assessment after their peak, will be censored at their last quantifiable assessment. Participants who stay unquantifiable during quarantine will be excluded from this analysis. The number of the excluded participants will be displayed.

In the case of one or more missing qRT PCR result in between two quantifiable PCR results, the duration will still be computed.

In the case of one or more missing qRT PCR measurements at the end of the period, not followed by any quantifiable result (i.e. without any available result or with only non-quantifiable ones), the exact timing of the end of the viral shedding is unknown and the exact duration cannot be computed.

- Duration of quantifiable influenza viral culture measurements in nasal samples from Day 1 (pm) up to Day 8 (am). Duration is defined as the time (hours) from first quantifiable until first confirmed unquantifiable assessment after their peak measure (after which no further virus is detected). Similar approach as for the duration of quantifiable qRT-PCR will be used.
- Time to peak as measured by graded daily symptom score system (from Day 1 [am] to the time of peak daily symptom score). The TSS is calculated at each day and at each 3 timepoints. Per participant, the first time with the highest daily TSS will be selected between all calculated TSS.
- Number (%) of participants with at least one single symptom scored grade 2 or higher at any time, from Day 1 (am) up to Day 8 (am).
- Number (%) of participants with at least one single symptom scored grade 2 or higher by time point, from Day 1 (am) up to Day 8 (am).


## **Statistical Analysis Plan**

- Number (%) of participants with lab-confirmed infection and fever (≥37.9°C). the derivation of the lab-confirmed infection is described the section 14.1.2.1 (RT-PCR-confirmed influenza infection).
- Total weight of mucus produced from Day 1 (am) up to Day 8 (am). The sum of mucus weight will be calculated by participant over the period.
- Total number of tissues used by participants from Day 1 (am) up to Day 8 (am). The sum of number of tissues will be calculated by participant over the period.
- Number (%) of participants with Laboratory-confirmed symptomatic influenza infection (community acquired), defined as:
  - o Self-reported influenza-like symptoms, AND
  - Community acquired (not challenge virus) laboratory-confirmed influenza infection PCR measurement and/or lateral flow positive, or other equivalent) reported on any occasion from discharge from quarantine up to Day 90 and/or up to Day 180 (±14 days).
- Pharmacokinetic (PK) parameters following CD388 administration will be determined as appropriate from the available data including: maximum plasma concentration ( $C_{max}$ ), time to maximum plasma concentration ( $T_{max}$ ), area under the plasma concentration-time curve from time 0 to time of last quantifiable sample ( $AUC_{0-t}$ ), and area under the plasma concentration-time curve from time 0 extrapolated to infinity ( $AUC_{0-\infty}$ ).
- CD388 concentrations in nasopharyngeal swabs: All collected parameters will be described by day/timepoint.
- Plasma concentration at specific time points, or PK parameters across dose arms, will be compared to viral or symptomatic endpoints in an effort to characterize the exposure response of CD388, and will be reported separately.
- Cytokine/chemokine levels may be explored in nasal samples, related to CD388 and infection: . All collected parameters will be described by day/timepoint.
  - Description will be presented by sub-groups (infected vs uninfected (definition in section 4.1.2.1 (RT-PCR-confirmed influenza infection) and symptomatic infected vs asymptomatic infected subjects (definition in section 4.1.2.1 (RT-PCR-confirmed symptomatic influenza infection)) for comparison.
- Cytokine/chemokine levels may be explored in serum samples, related to CD388 and infection: All collected parameters will be described by day/timepoint.
   Description will be presented by sub-groups (infected vs uninfected (definition in section 4.1.2.1 (RT-PCR-confirmed influenza infection) and symptomatic infected vs asymptomatic infected subjects (definition in section 4.1.2.1 (RT-PCR-confirmed symptomatic influenza infection)) for comparison.
- Viral resistance markers relevant for CD388. All collected parameters corresponding to viral resistance markers will be described by day/timepoint.


## 4.2 Safety endpoints

The safety and tolerability will be evaluated by the monitoring of the occurrence of AEs and SAEs, reactogenicity events (diary card), physical examinations, vital signs, 12-lead ECG, clinical laboratory results (haematology, biochemistry, coagulation, serology, cardiac enzymes, urinalysis, urine pregnancy test, thyroid function test), spirometry and concomitant medications.

Safety and tolerability will be assessed over the whole study period, up to EOS (planned on Day  $180 \pm 14$  days).

#### 4.2.1 Adverse events

Adverse events (solicited and unsolicited) will be coded using the latest available version of the Medical Dictionary for Regulatory Activities (MedDRA) and will be classified by MedDRA Preferred Term (PT) and System Organ Class (SOC).

A Treatment Emergent Adverse Event (TEAE) will be defined as any AE that started from the time of first study treatment dose administered to the participant until last study visit (Day 180).

Two categories of AE will be defined:

- Solicited AE: predefined events for which participants are specifically questioned and which are noted by participants in a participant diary (Erythema, swelling/induration, pain/tenderness)
- Unsolicited AE: any AEs observed by the participant or PI/investigator which are not pre-listed/on a symptom diary card.

For this study, 4 periods will be defined for solicited/unsolicited TEAE reporting:

- Period 1 between the intake of the first dose of the IMP on Day -5 until just before the challenge virus inoculation on Day 0 (Period 1),
- Period 2 from challenge virus inoculation until Day 8/Discharge from the quarantine unit
- Period 3 from Day 8/ discharge from the quarantine unit to Day 28 (±3 days)
- Period 4 from Day 28 (±3 days) until EOS (Day 180 ± 14 days).

Handling of missing or incomplete dates in the definition of treatment emergence and attribution between the 4 periods is provided in Section 6.4.1.1.

The relatedness of AE will be defined as follow:

- Unrelated = Not related and Unlikely related
- Related = possibly, probably and definitely related

The grading of the severity of the AEs will use the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Paediatric Adverse Events, Corrected Version 2.1 (July 2017).


## 4.2.2 Laboratory endpoints

The following clinical laboratory tests are to be performed on collected blood samples at screening, admission (Day -6), Day -1, Day 7, Day 17, Day 28, Day 60, Day 120 and Day 180:

- Biochemistry: sodium, potassium, glucose, albumin, chloride, bicarbonate, calcium, uric acid, total protein, creatinine, total, direct and indirect bilirubin, inorganic phosphate, blood urea nitrogen, C-reactive protein, gamma glutamyl transferase (GGT), alkaline phosphatase, alanine transaminase (ALT), lactate dehydrogenase (LDH), aspartate transaminase (AST) and urea.
- Haematology: platelet count, white blood cell count (absolute), white blood cell
  differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood
  cell count, reticulocyte count (% and absolute), haemoglobin, haematocrit, mean
  corpuscular volume, mean corpuscular haemoglobin, and mean corpuscular
  haemoglobin concentration.
- Coagulation: prothrombin time (PT), activated partial thromboplastin time (APTT)
- Urinalysis: colour, specific gravity, appearance, pH, presence of blood, glucose, leukocytes, ketones, nitrites, proteins, urobilinogen, bilirubin by dipstick. Microscopy, culture, and sensitivity examination will be performed if the dipstick yields abnormal results.

The laboratory values will be graded using Division of AIDS (DAIDS) will be used for grading.

## 4.2.3 Other safety endpoints

## 4.2.3.1 Physical examinations

Complete physical examinations will be conducted to include a full systemic assessment and will be performed according to the SoE.

Directed physical examinations will be conducted as deemed appropriate by the investigator and may include examination of the eyes, ears, nose, throat, and chest (via stethoscope).

Assessment and grading of any upper respiratory tract (URT) (nasal discharge, otitis, pharyngitis, sinus tenderness) and lower respiratory tract (LRT) symptoms (abnormal breath sounds externally [e.g., stridor, wheezing] and on chest auscultation [rhonchi, crepitations or other]) will be performed. Physician-reported assessments of viral challenge-related illness will be graded in accordance with its intensity and documented in the source data.

Following viral challenge, additional symptoms that are not available in the list of symptoms of the symptom diary card and are deemed to be clinically significant in the opinion of the investigator will be captured as an AE.

Following viral challenge all unexpected (in the opinion of the investigator) directed physical examination findings will be captured as AEs, along with all other occurrences that meet the criterion for an AE.

#### 4.2.3.2 Vital signs and temperature

Vital signs assessments will be recorded as follows:


## **Statistical Analysis Plan**

- Tympanic temperature will be recorded in degrees Celsius.).
- Heart rate (HR) will be recorded in beats per minute.
- Respiratory rate (RR): respirations will be counted and recorded as breaths per minute.
- Blood pressure (BP): systolic BP and diastolic BP will be measured in millimeters of mercury (mmHg); measurements will be made whilst the participant is in a supine position. Where possible, the same arm will be used for all measurements.
- Peripheral arterial oxygen saturation (SpO2%) will be assessed using pulse oximetry.

Study specific normal ranges are provided in Table 1. If a result is out of the normal range and meets the criteria for an AE, the severity of the AE will be determined based on the DAIDS Table (July 2017).

Table 1: Vital signs normal range

| Vital Signs | Lower<br>Limit | Higher<br>Limit | Units |
|---|---|---|---|
| Tympanic temperature (above 37.8 classed as pyrexia) | 35.5 37.8 | | °C |
| Oxygen saturation | Normal is ≥95 | | % |
| Respiratory rate | 10 | 20 | breaths per minute |
| Heart rate | 40 | 100 | beats per minute |
| Systolic BP | 90 | 140 | mmHg |
| Diastolic BP | 50 | 90 | mmHg |

Source: Protocol Appendix 4: Normal Ranges

## 4.2.3.3 12-lead electrocardiogram (ECG):

The following 12-lead ECG parameters will be performed at screening, admission (Day -6), Day -1, Day 7 and Day 180:

- Heart rate in beats per minute
- QRS, PR interval, QT, QTc in milliseconds

Study specific normal ranges are provided in Table 2

Table 2: ECG normal range

| ECG Parameters | Lower Limit | Higher Limit | Units |
|-------------------------|-------------|----------------|-------|
| Heart rate | 40 | 100 | bpm |
| QRS | 60 | 120 | ms |
| PR interval | 120 | 220 | ms |
| QT | 320 | 450 | ms |
| OT (5:1 :: (5) | 220 | <450 (females) | |
| QTc (Fridericia/Bazett) | 320 | <430 (males) | ms |


## **Statistical Analysis Plan**

## 4.2.3.4 Reactogenicity events (diary card)

Participants will be provided with the reactogenicity diary card to complete, once daily from Day -5 to Day -1. Participants will be asked to provide severity grade for the following items in the diary card:

- Redness (recorded in cm)
- Swelling (recorded in cm)
- Pain/tenderness (at the injection site)

The grading scale used to assess the local reactions of injectable products as reported in the reactogenicity diary has been adopted from the FDA Center for Biologics Evaluation and Research (CBER) guidelines on toxicity grading scales for healthy adult volunteers enrolled in preventative vaccine clinical trials. In the event a local reaction is reported as an (S)AE, the grading scale will be documented in the associated AE/SAE form by the investigator.

## **Local Reaction Grading Scale:**

| Local Reaction to<br>Injectable Product | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe (Grade<br>3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Pain | Does not interfere with activity | Repeated use of<br>non-narcotic pain<br>reliever > 24 hours<br>or interferes with<br>activity | Any use of narcotic pain reliever or prevents daily activity | Emergency room<br>(ER) visit or<br>hospitalization |
| Tenderness | Mild discomfort to touch | Discomfort with movement | Significant discomfort at rest | ER visit or hospitalization |
| Erythema/Redness <sup>a</sup> | 2.5 – 5 cm | 5.1 cm – 10 cm | >10 cm | Necrosis or exfoliative dermatitis |
| Induration/Swelling <sup>b</sup> | 2.5 – 5 cm and does<br>not interfere with<br>activity | 5.1 – 10 cm or interferes with activity | >10 cm or<br>prevents daily<br>activity | Necrosis |

#### 4.2.4 Concomitant medications

Concomitant medication data will be coded according to the latest available version of the WHO-Drug dictionary.

Concomitant medications are defined as any medication which was taken at any time on or after the start of study treatment, i.e:

- Started before or on first IMP intake and still ongoing at first IMP intake
- Started after first IMP intake


All other medications started and stopped before first IMP intake will be considered prior medications.

In case of missing start date, the medication should be assumed prior and concomitant unless the end data indicates was stopped prior to first IMP intake.

Handling of missing or incomplete dates is described in Section 6.4.1.1.

## 5 Statistical and Analytical Methods

#### 5.1 General considerations

The statistical analyses are performed in accordance with the ICH E9 guideline and other relevant guidance.

The statistical analyses will be performed by an external Contract Research Organisation (CRO), under the responsibility of the Sponsor.

#### 5.1.1 Presentation of results

The following descriptive statistics will be presented:

- For quantitative variables: number of available participants with the data point, number of missing data, mean, standard deviation (SD), median, Q1 (first quartile), Q3 (third quartile), minimum, and maximum values. When relevant, confidence intervals (CIs) will be computed for the mean (Student CI) and/or the median (Hahn & Meeker 1991).
- For qualitative variables: number of available participants with the data point, number
  of missing values, frequency counts for each category and corresponding percentage.
  Except if otherwise specified, percentages will be calculated using the number of
  available data as the denominator (i.e., not including missing values). When relevant,
  Cls will be computed. If not otherwise specified, the Clopper-Pearson method will be
  used to compute Cls for proportions.

## 5.1.2 Significance testing and estimation

#### 5.1.2.1 Between group comparisons:

For continuous variables (either raw data or log-transformed data) the difference in means, the standard error and the 95% 2-sided CI will be presented. In case of log-transformed variables, in addition to the previous statistics on the log-transformed data, the geometric means and geometric mean ratio and its 95% 2-sided CI for the original variable will be presented. The Wilcoxon rank-sum test will be used.

For categorical variables, differences in absolute frequency and/or relative risks will be presented, with their 95% 2-sided CIs. Except otherwise specified the Fisher exact test will be used to compare frequencies between study intervention arms

## 5.1.2.2 Control of overall type-I error:

Between-arm comparisons will be performed using appropriate hypothesis tests at the 2.5% 1-sided significance level, except if otherwise specified. No adjustment of the type-1 error rate for multiple comparisons will be done and each test will use a nominal level of 0.025 1-sided.


## 5.2 Sequence of analyses

A first interim analysis will be performed, by an unblinded team not involved in daily management of the study, for participants in Cohort 1 who have completed the inpatient phase at the time the interim analysis is performed. An optional second interim analysis may be performed by an unblinded team not involved in daily management of the study, within Cohort 2, depending on the outcome of the first interim analysis (See Figure 1 in section 2.3.1)

A final analysis (Day 180) is planned after all participants have completed the EOS (or early withdrawal) visit, after data management is complete and after the blind data review and database lock.

All statisticians/programmers except those involved in the interim analysis will remain blinded until the final DB lock. If SAP updates are necessary, they will be handled by this blinded team.

#### 5.3 Planned analysis

The lists of statistical Tables, Figures and Listings (TFL) are provided in Section 12.

## 5.3.1 Participant disposition and study discontinuations

Participant disposition will be described in a table (Statistical Table 14.1.1). The following variables will be tabulated:

- Number of randomized participants by randomised arm and overall
- Number of participants receiving IMP doses of CD388/placebo, by randomised arm and overall
- Number of participants receiving challenge virus, by randomised arm and overall

Analysis sets will be tabulated, overall and by randomised arm along with reasons for exclusion from the Enrolled, ITT, ITT-I, PP and SAF sets (Statistical Table 14.1.2). Individual data on the inclusion to/exclusion from each of the defined analysis sets will be provided in Listing 16.2.3.

Study duration and premature study discontinuation will be summarized using the following variables on the Enrolled Set, overall and by randomized arm:

- Number of participants who completed/discontinued the study, total and per treatment arm
- Reason for study discontinuation, total and per randomised arm
- Study duration defined as the difference between end of study date and date of enrolment +1, total and per randomised arm

The results will be included in Statistical Table 14.1.1.

Individual data on end of study information and reasons for discontinuation will be provided in Listing 16.2.1.

Visit dates (including date of consent) will be presented in Listing 16.2.4.10.

#### 5.3.2 Protocol deviations

All protocol deviations 3.1.13.1.2 will be summarized (number and percentage of subjects with at least one protocol deviation, with at least one minor deviation and at least one major 

deviation, and the number of major protocol deviations by deviation category) by randomised arm for the ITT set (Statistical Table 14.1.3). Individual data on protocol deviations will also be provided in Listing 16.2.2.

## 5.3.3 Demographics and baseline characteristics

The following demographics variables will be summarised by randomised arm on the ITT, ITT-I, PP and SAF analysis sets (Statistical Table 14.1.4.1 to .4) and individual data provided in Listing 16.2.4.1:

- Sex
- Age
- Ethnicity
- Race
- Weight
- Height
- BMI

The following baseline characteristics will be listed by treatment arm on the ITT set:

- Weight, height and BMI (Listing 16.2.4.2)
- Alcohol breath test and drugs of abuse and cotinine use (Listings 16.2.4.3 and 16.2.4.4)
- Urine pregnancy test, serum follicle-stimulating hormone (FSH) levels and serum betahuman chorionic gonadotrophin ( $\beta$ -HCG) pregnancy test (Listing 16.2.4.5)
- HIV, hepatitis B and C and thyroid function data will be presented in Listing 16.2.4.6

Eligibility criteria and randomisation information will be presented respectively in Listings 16.2.4.7 and 16.2.4.8.

Nasal swab respiratory pathogen screen data will be presented in Listing 16.2.4.11.

#### 5.3.4 Medical history – Prior medications

Medical history will be tabulated by SOC and PT by randomisation arm on the ITT set (Statistical Table 14.1.5). Note that the participant with the same System Organ Class /Preferred Term will be counted once.

Medical history for each participant will be reported in Listing 16.2.4.9.

Prior medications will be tabulated by ATC Level 2 code and Preferred Name by randomisation arm on ITT and PP set (Statistical Tables 14.1.6. and 14.1.6.2)

Prior medications for each participant will be reported in Listing 16.2.4.12 (together with concomitant medications).

#### 5.3.5 Concomitant medications

Concomitant medications will be tabulated on the ITT and PP by ATC Level 2 code and Preferred Name by randomised arm (Statistical Tables 14.1.7.1 and 14.1.7.2). Note that the participant with the same ATC Level 2/Preferred Name will be counted once.

Concomitant medications for each participant will be reported in Listing 16.2.4.12 (together with prior medications).


## 5.3.6 Spirometry

Spirometry will be performed according to hVIVO SOPs. Height at screening will be used as the baseline measurement for all spirometry assessments.

The following parameters will be performed at eligibility only (Spirometry may be repeated at any time in the event of respiratory signs or symptoms (repeated coughing, bradypnea, tachypnoea, rales, and rhonchi) or respiratory difficulties):

- FEV1 (observed and percent predicted)
- FVC (observed and percent predicted)
- FEV1/FVC (observed and percent predicted)

Study specific normal ranges are provided on Table 3

**Table 3: Spirometry normal range** 

| <b>Spirometry Parameters</b> | Lower Limit | Higher Limit |
|---|---|---|
| FEV <sub>1</sub> | Normal if ≥80% of the predicted value | |
| FEV <sub>1</sub> /FVC | Normal if ≥70% (≥0.7) of the predicted value | |

#### 5.3.7 Efficacy analyses

## **5.3.7.1** Primary efficacy analysis

## 5.3.7.1.1 Statistical hypotheses for primary efficacy analysis

The primary statistical hypothesis is that prophylactic treatment with CD388 at the dose of 150 mg will statistically significantly reduce influenza VL-AUC as determined by qRT-PCR on nasal samples compared to placebo. The second dose arm (50 mg) will also be compared to placebo, using a similar hypothesis.

Note that, as stated in Section 5.1.2, these two hypotheses will both be tested and compared to a one-sided type-1 error rate of 0.025, without adjustment.

The following statistical hypotheses will be tested:

- 1:  $H_{01}$ : AUC VL (150 mg)  $\geq$  AUC VL (Placebo) vs  $H_A1$ : AUC VL (150 mg) < AUC VL (Placebo)
- 2:  $H_{02}$ : AUC VL (50 mg)  $\geq$  AUC VL (Placebo) vs  $H_A2$ : AUC VL (50 mg) < AUC VL (Placebo)

## 5.3.7.1.2 <u>Statistical methods for primary efficacy analysis</u>

The primary efficacy endpoint is the total AUC of Influenza H3N2 A/Perth/16/2009 viral load measured by qRT-PCR on nasal samples.

Provided this is a phase IIa, proof of concept study, the primary scientific question is that of the prophylactic effect when treatment and viral challenge are administered as per protocol (efficacy) rather than that of the prophylactic effect in real life condition (effectiveness). Consequently, the primary efficacy analysis will be conducted on the PP analysis population.

Descriptive statistics for the mean and median and the 2-sided 95% CI for the mean will be presented by study arm. The significance of the difference between each CD388 arm and the


placebo arm will be analysed using the Wilcoxon rank-sum test. The estimator of the location shift in area under the curve (AUC), with 95% CI will be obtained via the Hodges-Lehman (+Moses) method. The one-sided p-value will be presented (Statistical Table 14.2.1.1).

Boxplots of the VL-AUC per randomized arm (Figure 14.2.1.1.1) and a plot of VL mean values over time per randomised arm (Figure 14.2.1.1.2) will be prepared.

Individual qRT-PCR data and VL-AUC for each participant will be reported respectively in the listings 16.2.6.1 and 16.2.6.4.

## 5.3.7.1.3 <u>Supplementary efficacy analyses for primary efficacy endpoint</u>

These supplementary analyses aim at documenting the influence of the choice of the analysis set on the results.

The same analyses methods as described in Section 5.3.7.1.2 for the PP analysis set and the same figures will be produced for the ITT (Statistical Table 14.2.1.2.1, Figures 14.2.1.2.1.1 and 14.2.1.2.1.2) and the ITT-I (Statistical Table 14.2.1.2.2, Figures 14.2.1.2.2.1 and 14.2.1.2.2.2) analysis sets.

## 5.3.7.2 Secondary efficacy analyses

Secondary efficacy analyses will be based on the PP analysis set only except if otherwise specified.

## 5.3.7.2.1 Virologic endpoints

Individual viral load data and derived efficacy response data for each participant by day/timepoint will be reported respectively in the listings 16.2.6.1 and 16.2.6.4.

Viral load from qRT-PCR and from viral culture will be described by day and by timepoint (respectively Statistical Tables 14.2.4.1 (PP), 14.2.4.2 (ITT), 14.2.4.3 (ITT-I) and Statistical Tables 14.2.8.1 (PP), 14.2.8.2 (ITT), 14.2.8.3 (ITT-I))

## 5.3.7.2.1.1 Peak viral load by qRT-PCR

The peak viral load of influenza from Day 1 (pm) up to Day 8 (am) will be presented by randomized arm using descriptive statistics for quantitative variables with 95% CI for the mean. The between mean difference and its 95% CI will be presented. The significance of the differences between each CD388 arm and the placebo arm will be analyzed using the Wilcoxon rank sum test. The one-sided p-values will be presented (Statistical Table 14.2.2.1). Boxplot of the Peak viral load for each randomized arm will be prepared (Figure 14.2.2.1).

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.2.2 and Figure 14.2.2.2).

## 5.3.7.2.1.2 Time to confirmed negative test by qRT-PCR

The Time (in hours) to confirmed negative test by qRT-PCR will be analysed using the Kaplan-Meier method. A Kaplan-Meier plot by randomized arm will be displayed showing the Time to confirmed negative test by qRT-PCR (with the time axis in hours since Day 1 (pm)). A table will accompany the plot and will display by randomised arm, the number of participants with event, the number of participants censored, the median, 25th percentile and 75th percentile of the time to confirmed negative test by qRT-PCR and their 95% confidence intervals. It will




## **Statistical Analysis Plan**

also display the Kaplan-Meier estimates of the cumulative proportion of subjects with an event (ie, with a negative qRT-PCR test) at specific time points in hours. The actual time of each assessment will be used in the calculation of Kaplan-Meier estimates. The significance of the difference between each CD388 arm and placebo will be analyzed using the Gehan-Wilcoxon test (one side p-value). The number of participants who do not have a detectable qRT-PCR value during quarantine excluded from the analysis will be also displayed. (Statistical Table 14.2.3.1) and Figure 14.2.3.1).

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.3.2 and Figure 14.2.3.2).

## 5.3.7.2.1.3 VL-AUC by viral culture

The VL-AUC will be computed on the viral culture results from nasal samples collected twice daily starting with the first day post-viral challenge (Day 1 pm) up to discharge from quarantine (Day 8).

The same analyses methods as described in Section 5.3.7.1.2 will be performed for the PP and the ITT-I analysis sets (Statistical Tables 14.2.5.1 and 14.2.5.2).

Boxplots of the VL-AUC per randomized arm (Figure 14.2.4.1.1 (PP) and 14.2.4.2.1 (ITT-I)) and a plot of VL mean values over time per randomized arm (Figure 14.2.4.1.2 (PP) and 14.2.4.2.2 (ITT-I)) will be prepared.

## 5.3.7.2.1.4 Peak viral load by viral culture

The peak viral load of influenza will be presented by randomized arm using descriptive statistics for quantitative variables with 95% CI for the mean. The between mean difference and its 95% CI will be presented. The significance of the difference between CD388 arm and placebo will be analysed using the Wilcoxon rank sum test. The one-sided p-value will be presented. (Statistical Table 14.2.6.1)

Boxplot of the Peak viral load by viral culture per randomized arm will be prepared (Figure 14.2.5.1).

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.6.2 and Figure 14.2.5.2).

#### 5.3.7.2.1.5 Time to confirmed negative test by viral culture

The Time (in hours) to confirmed negative test by quantifiable viral culture will be analysed using Kaplan-Meier method. A Kaplan-Meier plot by randomized arm will be displayed showing the Time to confirmed negative test by quantifiable viral culture (with the time axis in hours since Day 1 (pm)). A table will accompany the plot and will display by randomized arm, the number of participants with event, the number of participants censored, the median, 25th percentile and 75th percentile of the time to confirmed negative test by viral culture and their 95% confidence intervals. It will also display the Kaplan-Meier estimates of the cumulative proportion of subjects' event free with an event (ie, with a negative viral culture test) at specific time points by randomized arm in hours. The actual time of each assessment


will be used in the calculation of Kaplan-Meier estimates. The significance of the difference between each CD388 arm and placebo will be analyzed using the Gehan-Wilcoxon test (one sided p-value). The number of participants who do not have a detectable viral culture value during quarantine excluded from the analysis will be also displayed. (Statistical Table 14.2.7.1 and Figure 14.2.6.1).

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.7.2 and Figure 14.2.6.2).

## 5.3.7.2.1.6 Incidence of qRT-PCR-confirmed influenza infection

The incidence of qRT-PCR-confirmed influenza infection will be presented by randomized arm using descriptive statistics for qualitative variables with the 95% CI for the incidence. The significance of the difference between each CD388 arm and the placebo arm will be analysed using the Fisher's exact test with a one-sided alpha level of 0.025 (Statistical Table 14.2.14.1). This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.14.2).

## 5.3.7.2.1.7 Incidence of occurrence of at least 1 positive quantitative (≥LLOQ) cell culture

The occurrence of at least 1 positive quantitative (≥LLOQ) cell culture measurement in nasal samples, from Day 1 (pm) up to Day 8 (am) will be presented by randomized arm using descriptive statistics for qualitative variables with the 95% CI for the incidence. The significance of the difference between each CD388 arm and the placebo arm will be analysed using the Fisher's exact test with a one-sided alpha level of 0.025 (Statistical Table 14.2.15.1). This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.15.2).

#### 5.3.7.2.1.8 Incidence of qRT-PCR-confirmed symptomatic influenza infection

The incidence will be presented by randomized arm using descriptive statistics for qualitative variables with the 95% CI for the rate. The significance of the difference between each CD388 arm and the placebo arm will be analysed using the Fisher's exact test with a one-sided alpha level of 0.025 (Statistical Table 14.2.16.1).

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.16.2).

# 5.3.7.2.1.9 Incidence of qRT-PCR-confirmed moderately severe symptomatic influenza infection

The incidence will be presented by randomized arm using descriptive statistics for qualitative variables with the 95% CI for the rate. The significance of the difference between each CD388 arm and the placebo arm will be analysed using the Fisher's exact test with a one-sided alpha level of 0.025 (Statistical Table 14.2.17.1).

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.17.2).

#### 5.3.7.2.1.10 Culture lab-confirmed symptomatic influenza infection

The incidence will be presented by randomized arm using descriptive statistics for qualitative variables with the 95% CI for the rate. The significance of the difference between each CD388


arm and the placebo arm will be analysed using the Fisher's exact test with a one-sided alpha level of 0.025 (Statistical Table 14.2.18.1).

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.18.2).

## 5.3.7.2.2 Clinical symptoms

Individual and total clinical symptoms score and derived efficacy response data for each participant by day/timepoint will be reported respectively in the listings 16.2.6.2 and 16.2.6.4. The TSS will be described by day and by timepoint (Statistical Tables 14.2.13.1 (PP), 14.2.13.2 (ITT) and 14.2.13.3 (ITT-I).

## 5.3.7.2.2.1 Area under the curve over time of total clinical symptoms score (TSS-AUC)

The TSS-AUC collected from Day 1 (am) up to Day 8 (am) will be presented by randomized arm using descriptive statistics for quantitative variables with 95% CI for the mean. The between mean difference and its 95% CI will be presented. The significance of the difference between each CD388 arm and the placebo arm will be analysed using the Wilcoxon rank sum test. The one-sided p-value will be presented (Statistical Table 14.2.9.1).

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.9.2).

Boxplots of the TSS-AUC per randomized arm (Figure 14.2.7.1.1 (PP) and 14.2.7.2.1 (ITT-I)) and a plot of TSS mean values over time per randomised arm (Figure 14.2.7.1.2 (PP) and 14.2.7.2.2 (ITT-I)) will be prepared.

#### 5.3.7.2.2.2 Peak of total clinical symptoms score

The peak of TSS will be presented by randomized arm using descriptive statistics for quantitative variables with 95% CI for the mean. The between mean difference and its 95% CI will be presented. The significance of the difference between CD388 arm and placebo will be analysed using the Wilcoxon rank sum test. The one-sided p-value will be presented. (Statistical Table 14.2.10.1)

Boxplot of Peak total clinical symptoms score per randomised arm will be prepared (Figure 14.2.8.1).

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.10.2 and Figure 14.2.8.2).

#### 5.3.7.2.2.3 Individual peak daily total clinical symptoms score

The individual peak daily TSS from Day 1 up to Day 8 will be presented by randomized arm using descriptive statistics by day for quantitative variables with 95% CI for the mean. The between mean difference and its 95% CI will be presented. The significance of the difference between CD388 arm and placebo will be analysed using the Wilcoxon rank sum test. The one-sided p-value will be presented. (Statistical Table 14.2.11.1)

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.11.2).


A plot of peak daily TSS mean values over time per randomised arm (Figure 14.2.9.1 (PP) and 14.2.9.2 (ITT-I)) will be prepared.

## 5.3.7.2.2.4 Time to symptom resolution

The Time to symptom resolution will be analysed using the Kaplan-Meier method. A Kaplan-Meier plot by randomised arm will be displayed showing the Time to symptom resolution (with the time axis as hours since peak daily symptom score). A table will accompany the plot and will display by randomized arm, the number of participants with event, the number of participants censored, the median, 25th percentile and 75th percentile of the time to symptom resolution and their 95% confidence intervals. It will also display the Kaplan-Meier estimates of the cumulative proportion of subjects' event free with an event (ie, with symptom resolution) at specific time points by randomized arm in hours. The actual time of each assessment will be used in the calculation of Kaplan-Meier estimates. The significance of the difference between each CD388 arm and placebo will be analyzed using the Gehan-Wilcoxon test (one sided p-value) (Statistical Table 14.2.12.1 and Figure 14.2.10.1).

This analysis will be repeated on the ITT-I analysis set (Statistical Table 14.2.12.2 and Figure 14.2.10.2).

#### 5.3.7.3 Tertiary/exploratory efficacy analyses

No inferential statistics will be computed for tertiary/exploratory efficacy endpoints. Their analyses will be only descriptive on PP analysis set.

Other tertiary/exploratory efficacy analyses may be conducted and will be described in a SAP amendment.

## 5.3.7.3.1 Quantitative tertiary/exploratory endpoints

Descriptive statistics for quantitative variables, including the 95% CI for the mean, will be tabulated for:

- Duration of quantifiable influenza qRT-PCR measurements in nasal samples from Day 1 (pm) up to Day 8 (am). (Statistical Table 14.2.19).
- Duration of quantitative influenza viral culture measurements in nasal samples from Day 1 (pm) up to Day 8 (am). (Statistical Table 14.2.20).
- Time to peak as measured by graded daily symptom score system (from Day 1 (am) to the time of peak daily symptom score). (Statistical Table 14.2.21).
- Total weight of mucus produced from Day 1 (am) up to Day 8 (am) (Statistical Table 14.2.22).
- Total number of tissues used by participants from Day 1 (am) up to Day 8 (am) (Statistical Table 14.2.23).
- Cytokine/chemokine levels may be explored in nasal samples, related to CD388 and infection. (Statistical Table 14.2.28.1 overall, by sub-groups 16.2.28.2 and 16.2.28.3 and listing 16.2.6.5)


• Cytokine/chemokine levels may be explored in serum samples, related to CD388 and infection. (Statistical Table 14.2.29.1 overall, by sub-groups 16.2.29.2 and 16.2.29.3 and listing 16.2.6.5)

#### 5.3.7.3.2 Qualitative tertiary/exploratory endpoints

Descriptive statistics for qualitative variables, including the 95% CI for the rates, will be tabulated for:

- Number (%) of participants with symptom scored grade 2 or higher, from Day 1 (am) up to Day 8 (am) (Statistical Table 14.2.24).
- Number (%) of participants with symptom scored grade 2 or higher by time point, from Day 1 (am) up to Day 8 (am) (Statistical Table 14.2.25).
- Number (%) of participants with lab-confirmed infection and fever (≥37.9°C) (Statistical Table 14.2.26).
- Number (%) of participants with Laboratory-confirmed symptomatic influenza infection (community acquired) (Statistical Table 14.2.27), defined as:
  - Self-reported influenza-like symptoms, AND
  - Community acquired (not challenge virus) laboratory-confirmed influenza infection PCR measurement and/or lateral flow positive, or other equivalent) reported on any occasion from discharge from quarantine up to Day 90 and/or up to Day 180 (±14 days).
- Viral resistance markers relevant for CD388. (Statistical Table 14.2.30 and listing 16.2.6.6)

#### 5.3.7.4 Other efficacy variables

The following data will be presented in listings on the ITT analysis set:

- Nasopharyngeal swab for rapid viral antigen test at discharge from quarantine (Listing 16.2.6.7)
- 24-hour tissue count and nasal discharge weight (Listing 16.2.6.3)
- Blood Serum anti-drug antibodies (ADA) will be presented by randomized arm by day in term of presence/absence of ADA (Statistical table 14.2.31.1) and in term of titer levels (Statistical table 14.2.31.2) and Listing 16.2.6.8.

#### 5.3.8 Safety analyses

Safety variables will be tabulated and presented for all participants included in the Safety analysis set (SAF).

#### 5.3.8.1 Extent of exposure and compliance

Compliance with IMP (CD388/placebo) will be computed on the ITT and SAF set by randomized arm (Statistical Tables 14.1.8.1 and 14.1.8.2) by assessing the proportion of participants actually receiving a full dose of IMP as prescribed.


IMP/ Placebo dosing and Challenge virus inoculation information for each participant will be reported respectively in Listings 16.2.5.1 and 16.2.5.2.

#### 5.3.8.2 Adverse events

#### 5.3.8.2.1 Adverse event tabulations:

Tabulation of solicited or unsolicited AEs will be done according to four periods based on their date and time of start, as presented in Table 4:

Table 4: periods for AE tabulation

| Period | Description | from | to |
|---|---|---|---|
| Period 1 | Treatment Emergent/ Pre-viral Challenge Emergent Adverse Events | First intake of IMP on Day -5 | Just before challenge virus inoculation on Day 0 |
| Period 2 | Treatment and Viral Challenge<br>Emergent Adverse Events | Challenge virus inoculation on Day 0 | Actual discharge from the quarantine unit (as scheduled on Day 8 or later on PI's decision) |
| Period 3 | Post quarantine Adverse Events | Actual discharge from the quarantine unit | Day 28 (±3 days) |
| Period 4 | Post Day 28 Adverse Events | Day 28 | Day 180 (±14 days) (EOS visit) |

Tabulation of adverse events will present the following information: number of participants with at least one occurrence of the event, corresponding percentage and number of events (if relevant).

The following tables will be produced by treatment arm (as treated):

#### 5.3.8.2.1.1 Summary table of adverse events (Statistical Table 14.3.1):

- Any AE
- Any TEAE (solicited + unsolicited TEAE)
- Any solicited AE during Period 1
- Any unsolicited TEAE across all periods (i.e. period 1, 2, 3 or 4)
- Any unsolicited TEAE during Period 1
- Any unsolicited TEAE during Period 1 and Period 2
- Any unsolicited TEAE during Period 2
- Any unsolicited TEAE during Period 2 and Period 3
- Any unsolicited TEAE during Period 3
- Any unsolicited TEAE during Period 3 and Period 4
- Any unsolicited TEAE during Period 4
- Any unsolicited TEAE during Period 1 leading to study treatment discontinuation (only relevant for Period 1)


## **Statistical Analysis Plan**

- Any unsolicited TEAE across all periods (i.e. period 1, 2, 3 or 4) leading to study discontinuation
- Any unsolicited TEAE during Period 1 leading to study discontinuation
- Any unsolicited TEAE during Period 1 and Period 2 leading to study discontinuation
- Any unsolicited TEAE during Period 2 leading to study discontinuation
- Any unsolicited TEAE during Period 2 and Period 3 leading to study discontinuation
- Any unsolicited TEAE during Period 3 leading to study discontinuation
- Any unsolicited TEAE during Period 3 and Period 4 leading to study discontinuation
- Any unsolicited TEAE during Period 4 leading to study discontinuation
- Any unsolicited TEAE across all periods (i.e. period 1, 2, 3 or 4) considered related to the study treatment (at least possibly related)
- Any unsolicited TEAE during Period 1 considered related to the study treatment (at least possibly related)
- Any unsolicited TEAE during Period 1 and Period 2 considered related to the study treatment (at least possibly related)
- Any unsolicited TEAE during Period 2 considered related to the study treatment (at least possibly related)
- Any unsolicited TEAE during Period 2 and Period 3 considered related to the study treatment (at least possibly related)
- Any unsolicited TEAE during Period 3 considered related to the study treatment (at least possibly related)
- Any unsolicited TEAE during Period 3 and Period 4 considered related to the study treatment (at least possibly related)
- Any unsolicited TEAE during Period 4 considered related to the study treatment (at least possibly related)
- Any serious adverse events (SAE) across all periods (i.e. period 1, 2, 3 or 4)
- Any SAE during Period 1
- Any SAE during Period 1 and Period 2
- Any SAE during Period 2
- Any SAE during Period 2 and Period 3
- Any SAE during Period 3
- Any SAE during Period 3 and Period 4
- Any SAE during Period 4
- Any TESAE leading to study treatment discontinuation, across all periods (i.e. period 1, 2, 3 or 4).
- Any TESAE leading to study discontinuation, across all periods (i.e. period 1, 2, 3 or 4)
- Any SAE considered related to the study treatment, across all periods (i.e. period 1, 2, 3 or 4)
- Death (if any)


## **Statistical Analysis Plan**

#### 5.3.8.2.1.2 Detailed Tables:

- Any solicited AE by PT during Period 1 (Statistical Table 14.3.2.1)
- Any unsolicited TEAE by SOC and PT
  - o across all periods (i.e. period 1, 2, 3 or 4) (Statistical Table 14.3.2.2)
  - Period 1 (Statistical Table 14.3.2.3)
  - Period 1 and Period 2 (Statistical Table 14.3.2.4)
  - o Period 2 (Statistical Table 14.3.2.5)
  - Period 2 and Period 3 (Statistical Table 14.3.2.6)
  - Period 3 (Statistical Table 14.3.2.7)
  - o Period 3 and Period 4 (Statistical Table 14.3.2.8)
- Any unsolicited TEAE by SOC, PT and relatedness
  - o Across all periods (i.e. period 1, 2, 3 or 4) (Statistical Table 14.3.3.1)
  - o Period 1 (Statistical Table 14.3.3.2)
  - Period 1 and Period 2 (Statistical Table 14.3.3.3)
  - Period 2 (Statistical Table 14.3.3.4)
  - Period 2 and Period 3 (Statistical Table 14.3.3.5)
  - Period 3 (Statistical Table 14.3.3.6)
  - Period 3 and Period 4 (Statistical Table 14.3.3.7)
- Any solicited AE by PT and maximum severity during Period 1 (Statistical Table 14.3.4.1)
- Any unsolicited TEAE by SOC/PT and maximum severity
  - Across all periods (i.e. period 1, 2, 3 or 4) (Statistical Table 14.3.4.2)
  - Period 1 (Statistical Table 14.3.4.3)
  - Period 1 and Period 2 (Statistical Table 14.3.4.4)
  - Period 2 (Statistical Table 14.3.4.5)
  - o Period 2 and Period 3 (Statistical Table 14.3.4.6)
  - Period 3 (Statistical Table 14.3.4.7)
  - Period 3 and Period 4 (Statistical Table 14.3.4.8)
- All unsolicited TEAE leading to study treatment discontinuation, by SOC and PT during Period 1 (only relevant for Period 1) (Statistical Table 14.3.5)


- Any unsolicited TEAE leading to study discontinuation, across all periods (i.e. period 1, 2, 3 or 4), by SOC and PT (Statistical Table 14.3.6)
- All unsolicited TESAEs by SOC and PT across all periods (i.e. period 1, 2, 3 or 4) (Statistical Table 14.3.7.1)
- Any SAE by SOC and PT
  - o Period 1 (Statistical Table 14.3.7.2)
  - o Period 1 and Period 2 (Statistical Table 14.3.7.3)
  - Period 2 (Statistical Table 14.3.7.4)
  - o Period 2 and Period 3 (Statistical Table 14.3.7.5)
  - Period 3 (Statistical Table 14.3.7.6)
  - Period 3 and Period 4 (Statistical Table 14.3.7.7)
- Any SAE by SOC, PT and relatedness across all periods (i.e. period 1, 2, 3 or 4) (Statistical Table 14.3.8)

#### 5.3.8.2.2 Adverse event listings:

A by-participant AE data listing including participant identifier, onset and resolution dates, relative study days based on date of first dose IMP/Placebo (for start and end date of AE, duration of AE), period, verbatim term, system organ class, preferred term, treatment, severity, relationship to treatment, action taken, and outcome will be provided:

- For solicited Adverse events in listing 16.2.7.1.1
- For unsolicited Adverse Events in Listing 16.2.7.1.2
- For unsolicited Serious Adverse Events in Listing 16.2.7.1.3
- For unsolicited treatment related TEAES in Listing 16.2.7.1.4
- For unsolicited AE leading to study discontinuation in Listing 16.2.7.1.5
- For Deaths (if any) Listing 16.2.7.1.6

#### 5.3.8.3 Laboratory safety variables

The laboratory data will be directly transferred from the central laboratory to the data management department. Any clinically significant change occurring during the trial must be recorded as an Adverse Event in the CRF.

Laboratory evaluations will be summarised by visit and by treatment arm on the SAF analysis set.

For each biochemistry, haematology and coagulation variable:

Quantitative descriptive statistics will be tabulated at each time point over the course
of the study (e.g., at each visit) on raw values and change from baseline (Statistical
Table 14.3.9.1.1 and 14.3.9.1.2)

Shift tables will be presented to show the number of subjects with each toxicity grade (1,2,3, or 4/5) at baseline versus each post-baseline visit and the worst post-baseline grade (including any unscheduled visits). For those laboratory parameters for which high toxicity grades are specified for both low and high values (e.g., sodium, potassium), shifts in toxicity will be presented for high and low toxicities separately. The percentages will be based on the number


of subjects with both a baseline and post-baseline (at the specified visit) assessment of the specific laboratory parameter. For parameters which can not be graded with DAIDS, shift tables will be presented using investigator's interpretation (normal, abnormal NCS and abnormal CS (Statistical Table 14.3.9.2)The number and percentage of subjects with at least a 2-grade increase from baseline at any post-baseline study visit, including unscheduled visits, will be summarized by laboratory parameter and treatment group. Percentages for each lab test will be based on the number of subjects with both a baseline and a post-baseline evaluation of the particular laboratory test(Statistical Table 14.3.9.3)Plots of mean raw values of each biochemistry, haematology and coagulation parameters over time per randomized arm will be produced (Statistical Figures 14.3.1).

All urinalysis parameters will also be tabulated as qualitative and/or quantitative variables (Statistical table 14.3.9.4)

All laboratory results will be presented in Listings 16.2.8.1 to .4.

The following listings will be presented:

- Biochemistry
- Biochemistry all results for subjects who have at least one 2-grade increase in a biochemistry parameter
- Haematology
- Haematology all results for subjects who have at least one 2-grade increase in a hematology parameter
- Urinalysis
- Coagulation

#### 5.3.8.4 Physical examinations

All individual data for complete and direct physical examination will be provided respectively in Listing 16.2.9.

#### 5.3.8.5 Vital signs and tympanic temperature

- Quantitative descriptive statistics (Raw values and change from baseline) will be tabulated by treatment arm for each vital sign recorded (tympanic temperature, heart rate, respiratory rate, systolic and diastolic blood pressure and peripheral arterial oxygen saturation) at each time point over the course of the study (Statistical Table 14.3.10.1 for Raw values and 14.3.10.2 for Change from baseline).
- Qualitative descriptive statistics (normal/abnormal (outside of normal range)) will be presented for each vital sign at each time point over the course of the study by randomised arm (Statistical Table 14.3.10.3).
- All individual measurements will be provided in Listing 16.2.10

#### 5.3.8.6 12-Lead Electrocardiogram

• Quantitative descriptive statistics (Raw values and change from baseline) will be tabulated by treatment arm for each 12-Lead ECG parameters recorded (Heart rate,




QRS, PR interval, QT, QTc) at each time point over the course of the study (Statistical Tables 14.3.11.1.1 and 14.3.11.1.2).

- Qualitative descriptive statistics (normal/abnormal (outside of normal range)) will be presented for each 12-ead ECG parameters at each time point over the course of the study by treatment arm (Statistical Table 14.3.11.2).
- All individual measurements will be provided in Listing 16.2.11

#### 5.3.8.7 Spirometry

All individual data for spirometry will be provided in Listing 16.2.12.

#### 5.3.8.8 Reactogenicity events (diary card)

All individual data for reactogenicity events will be provided in Listing 16.2.13.

#### 5.3.8.9 Concomitant medications

Concomitant medications will be presented by ATC class level 2 and Preferred Name by treatment arm (Statistical Table 14.1.7).

Individual data on previous and concomitant medications for each participant will be reported in Listing 16.2.4.12.

#### 6 Data handling conventions

#### **6.1 Definitions**

#### 6.1.1 Baseline definition

For this study, the definition of a baseline value is only needed for the computation of changes for baseline for safety endpoints.

The baseline is defined as the last non-missing observation prior to the administration of the dose of study IMP will be used as the baseline value. This will usually correspond to the measurement performed at the admission visit on Day -6 or a re-test performed thereafter but before IMP administration on Day -5. In case of missing value at Day -5, the last available value recorded during the screening period will be used as the baseline value.

If all pre-dose/pre-challenge measurements are missing then baseline will be considered as missing, and no change from baseline and no percentage change from baseline will be computed.

#### 6.1.2 Quarantine discharge

Unless otherwise specified, Quarantine Discharge refers to the actual quarantine discharge day regardless of whether discharge from quarantine occurred as scheduled on Day 8, or later following the PI's decision to extend the quarantine period for a given participant.


#### 6.2 Retest, Outliers

#### 6.2.1 Retests

The retests will be managed as follow:

- Any retest before first IMP administration: the last available value before first IMP administration will be used as the baseline (see Section 6.1.1)
- Any other retest: Retest values will not be used in statistical analyses except if otherwise specified during the data review meeting. All available values (including retest values) will be presented in the data listings.

#### 6.2.2 Outliers

All available data points will be included in the analyses, unless a clear reason is available to exclude a given data point. Consequently, all potential outlier data will be reviewed during the Blinded Data Review Meeting (BDRM) and decisions regarding their use in the statistical analyses will be made.

#### 6.3 Visit windows, unscheduled visits

#### 6.3.1 Windows for time points

All visits will be analysed as entered in the database except if otherwise specified during the data-review meeting.

#### 6.3.2 Unscheduled visits

Unscheduled visit measurements may be used to provide a measurement for a baseline or endpoint value if appropriate according to their definition. Other unscheduled visits data will not be analysed, but corresponding data will be presented in the individual data listings and any relevant safety data will be described in the CSR.

#### 6.4 Missing data and analysis rules

In the presence of missing data, analysis rules are described in the following sections. In case of specific cases, data will be reviewed during the BDRM and decisions to derive the considered endpoint and how to derive it, will be documented in the BDRM minutes. If necessary, the SAP will be updated accordingly.

#### 6.4.1 Missing data

#### 6.4.1.1 Missing or incomplete dates:

For calculation / sorting / assignation based on dates (e.g. treatment emergent AEs, assignation of AEs between periods, concomitant medications, etc.), the following rules will apply:

• In case of AE with missing start date, it could be included in different analysis periods at the same time. If the AE could have started in multiple periods based on all the available information, it will be analysed in all the possible periods (i.e; for an AE with complete missing start date and end date after Day 28, the AE will belong to the 4 periods, for an AE with only the information that the AE started the month of treatment start and inoculation but before the Day 28, the AE will belong to period 1,


## **Statistical Analysis Plan**

2 and period 3). In case of partial date without ambiguity on the period, the date will be imputed by the first day of the month. In case of partial date without ambiguity on the period, the date will be imputed by the first month of the year.

- Medication with missing start date will be assumed prior and concomitant medication unless the end date indicates was stopped prior to first IMP intake.
- Medical history or disease diagnosis with missing/incomplete date will be assumed to have occurred before any study treatment except when the partial onset date or other available data indicates differently.

#### 6.4.1.2 Missing Viral Load and Total Symptom Score data

Missing Viral Load and Total Symptom Score data may impact the derivation of some of the study endpoints (AUC, sum of TSS, peak). General rules on how to derive these endpoints in the presence of missing data are provided in Section 7.

#### 6.4.1.3 Other missing data

No other missing data will be imputed except if otherwise specified in the SAP. Any other mechanisms to handle missing data will be outlined within the relevant endpoints section.

#### 6.4.2 Analysis rules

Except if otherwise specified, any data recorded as Detected, Not detected, Invalid, N/A or NDA will be presented as such in listings but will be replaced with the Assigned value described in the following table:

Table 5: Rules for handling qRT-PCR viral load, Viral culture results and HAI serology levels

| | | Assay Re | porting |
|---|---|---|---|
| Analysis | Assay | Reported result | Assigned value |
| | | Value | Use reported value |
| | Influenza Viral Culture assay | DETECTED | 1.0 TCID <sub>50</sub> /mL |
| Influenza titre | (TCID <sub>50</sub> /mL assay) | NOT DETECTED | 0.5 TCID <sub>50</sub> /mL |
| | (TCID50/IIIL assay) | INVALID | Missing data point |
| | | N/A | Missing data point |
| | | Value | Use reported value |
| | ant non | DETECTED | 1.94 Log <sub>10</sub> Copies/mL |
| PANFLU Viral Load | qRT-PCR<br>(Log10 copies/mL) | NOT DETECTED | 0.97 Log <sub>10</sub> Copies/mL |
| | (Log10 copies/IIIL) | INVALID | Missing data point |
| | | N/A | Missing data point |
| Influence costiled by | Influenza Neutralisation Assay | Value | Use reported value |
| Influenza antibody<br>titre | (virus focus reduction | NDA | 5 |
| uue | neutralisation | INVALID | Missing data point |
| | assay) | N/A | Missing data point |

N/A, not applicable; NDA, no detectable antibody




# **Statistical Analysis Plan**

Samples with titres above the assay ULOQ may be pre-diluted to obtain a quantifiable result and corrected for the dilution used, where possible.

#### 7 Derived data

| Derived variable | Derivation algorithm |
|---|---|
| Change from baseline to visit V | Change from baseline of variable X: |
| (continuous) | $X(Visit\ V) - X(baseline)$ |
| | <ul> <li>Negative values indicate a decrease in X</li> </ul> |
| | o Positive values indicate an increase in X |
| Event Duration (in days) | $(End\ date) - (Start\ date) + 1$ |
| Total symptom score | The TSS computation is based on the diary cards that participants complete 3 times per day from Day -1 to Day 7 and once on Day 8. |
| | At each assessment, the participants provide scores from 0 to 3 for a list of 13 symptoms (Runny nose, Stuffy nose, Sneezing, Sore throat, Earache, Malaise/tiredness, Headache, Muscle and/or joint ache, Chilliness/Feverishness, Cough, chest tightness, shortness of breath and wheeze), resulting in possible values from 0 to 39 for the TSS. |
| | An individual TSS is derived at each assessment of the diary card as the sum of the scores given to the 13 symptoms on that symptom score card. |
| | Handling of missing data for TSS calculations: If scores are missing for two or less symptoms within an otherwise completed diary card it will be assumed that the symptom(s) was(were) not present and as such a score of 0 will be given for that(/these) symptom(s) and the TSS endpoint derived as the sum of the available item scores. |
| | If more than two symptoms have not been completed for a specific assessment this will be treated as missing and no score will be derived for the TSS at that timepoint. |
| Area Under the Curve (AUC) of | Calculated using the trapezium rule [3]: |
| Viral Load and Total Symptom<br>Score | With n+1 measurements $y_i$ at times $t_i$ , (I = 0,.n), the AUC is calculated as: |
| (in log10 copies/mL * day for VL AUC) | $AUC = \frac{1}{2} \sum_{i=0}^{n-1} (t_{i+1} - t_i) (y_i + y_{i+1})$ |
| (in points * day for TSS AUC) | The actual time of each assessment will be used in the calculation. |
| | For VL AUC, 14 measurements are used for the computation (1 on Day 1, 2 on each day from Day 2 to Day 7 and 1 on Day 8). For TSS AUC, 22 measurements are used (3 on each day from Day 1 to Day 7 and 1 on Day 8). |
| | Handling of missing data for AUC calculations: |
| | The AUC calculation will be based on the available non-missing assessment values between the start and end of the defined AUC time period (Day 1 pm to Day 8 am for viral load, Day 1 am to Day 8 am for TSS) with the following exceptions: |
| | <ul> <li>If the first measurement or the last measurement of the AUC<br/>time period is missing, the following rules will be applied: In case</li> </ul> |




## Statistical Analysis Plan

| Derived variable | Derivation algorithm |
|---|---|
| | of the missing last measurement, the method of LOCF will be used. In case of the missing first measurement, the non missing first measurement will be reported at all missing measurement before. |
| | <ul> <li>Even if the formula above can still be calculated, too many<br/>missing measurements other than the first or last will impact the<br/>precision of the AUC for the given participant. As a general rule,<br/>the participant must have at least 1 non-missing data recording<br/>on each day between the start and end of the defined AUC time<br/>period to compute the AUC.</li> </ul> |
| | <ul> <li>Each specific case will be reviewed during the BDRM and<br/>decisions with their rationale documented in the BDRM minutes.</li> </ul> |
| Peak Viral Load<br>(or Peak Total Symptom score) | Computed as the maximum observed value for VL or TSS over the defined time period (D1 to D8) |
| | Handling of missing data for peak value calculation: In the presence of missing data, the maximum of the available data can still be identified, but it may not correspond to the true peak for the participant, when the peak would have corresponded to one of the missing assessments. |
| | Each specific case will be reviewed during the BDRM and decisions to derive a peak value and which value to use, with their rationale documented in the BDRM minutes. |

#### 8 Interim analysis

A first interim analysis will be performed, by an unblinded team not involved in daily management of the study, for participants in Cohort 1 who have completed the inpatient phase at the time the interim analysis is performed. An optional second interim analysis may be performed by an unblinded team not involved in daily management of the study, within Cohort 2, depending on the outcome of the first interim analysis

The following tables/figures will be produced at each interim analysis on PP population:

- Participant disposition (Statistical Table 14.1.1)
- Demographics and baseline characteristics PP analysis set (Statistical Table 14.1.4.3)
- Demographics and baseline characteristics SAF analysis set (Statistical Table 14.1.4.4)
- Primary efficacy analysis Area under the viral load-time curve (VL-AUC) from qRT-PCR (Statistical Table 14.2.1.1 and Figures 14.2.1.1.1 and 14.2.1.1.2)
- Peak viral load from qRT-PCR (Statistical Table 14.2.2.1 and Figure 14.2.2.1)
- Time to confirmed negative test by qRT-PCR (statistical Table 14.2.3.1 and Figure 14.2.3.1)
- Area under the curve over time of total clinical symptoms score (TSS-AUC) (Statistical Table 14.2.9.1 and Figures 14.2.7.1.1, 14.2.7.1.2)
- Peak of total clinical symptoms score (TSS) (Statistical Table 14.2.10.1 and figure 14.2.8.1)


- Time to symptom resolution (statistical Table 14.2.12.1 and Figure 14.2.10.1)
- Incidence of confirmed influenza infection by qRT-PCR (Statistical Table 14.2.14.1)
- Incidence of qRT-PCR-confirmed symptomatic influenza infection (Statistical Table 14.2.16.1)
- Incidence of qRT-PCR-confirmed moderately severe symptomatic influenza infection (Statistical Table 14.2.17.1)

The following tables/listings will be produced at each interim analysis on SAF population:

- Summary of adverse events (Statistical Table 14.3.1)
- Any unsolicited TEAE across all periods by SOC, PT and relatedness (Statistical Table 14.3.3.1)\*
- Any solicited AE by SOC/PT and maximum severity during Period 1 (Statistical Table 14.3.4.1)\*
- \* Tables will be produced in case if at least 20 reported adverse events in the database.
  - Solicited adverse events (Listing 16.2.7.1.1)
  - Unsolicited adverse events (Listing 16.2.7.1.2)
  - Reactogenicity events (Listing 16.2.13)

In the listings the participant numbers should be scrambled.

## 9 Statistical/Analytical issues

This section systematically reviews the topics listed in Section 11.4.2 of the ICH E3 guidance the ICH E3 as important features of the analysis, to ensure none of these topics has been overlooked in the current SAP and to facilitate the writing of the corresponding section in the CSR.

#### 9.1 Adjustments for Covariates

No adjustment for demographic or baseline measurements, or any other covariate are planned.

#### 9.2 Handling of Dropouts or missing data

Methods for handling missing data are described in Section 6.4.1.

#### 9.3 Interim Analyses and Data Monitoring

The interim analysis is described in Section 8.

#### 9.4 Multicentre studies

Not applicable: single centre study.

#### 9.5 Multiple Comparison/Multiplicity

See Section 5.1.2.2: as the study is of exploratory purpose, no adjustment for multiple comparisons / multiplicity of endpoints will be performed.




## 9.6 Use of an "Efficacy Subset" of Participants

Two subsets of the ITT efficacy set have been defined: the Intent-to-treat Infected (ITT-I) set and the Per Protocol (PP) set (see Section 3.3 for details).

#### 9.7 Active-Control Studies Intended to Show Equivalence

Not applicable.

#### 9.8 Examination of Subgroups

No specific subgroup analysis will be performed.

## 10 Modifications from the statistical section of the protocol

Not applicable

#### 11 Software documentation

All summaries and statistical analyses will be generated using SAS version 9.4 or higher.




# **Statistical Analysis Plan**

# 12 Tables, Figures and Listings

#### 12.1 List of tables

The list of tables is described in a separate document with mocks tables.

## 12.2 List of figures

The list of figures is described in a separate document with mocks figures.

## 12.3 List of listings

| n° | |
|---|---|
| 16.2.1 | End of study information / Discontinuation |
| 16.2.2 | Protocol deviations |
| 16.2.3 | Analysis sets membership and reasons for exclusion |
| 16.2.4 | Demographics and Baseline characteristics data |
| 16.2.4.1 | Demographic characteristics |
| 16.2.4.2 | Weight, Height and BMI |
| 16.2.4.3 | Alcohol breath test |
| 16.2.4.4 | Drugs of abuse and Cotinine use |
| 16.2.4.5 | Urine pregnancy test, serum FSH and β-HCG pregnancy test |
| 16.2.4.6 | HIV, Hepatitis B & C and Thyroid function |
| 16.2.4.7 | Eligibility criteria |
| 16.2.4.8 | Randomisation |
| 16.2.4.9 | Medical History |
| 16.2.4.10 | Visit dates |
| 16.2.4.11 | Nasal Swab for respiratory Pathogen Screen data |
| 16.2.4.12 | Prior and Concomitant Medication |
| 16.2.5 | Compliance and/or Drug Concentration Data |
| 16.2.5.1 | IMP/ Placebo dosing |
| 16.2.5.2 | Challenge virus Inoculation |
| 16.2.6 | Individual Efficacy Response Data |
| 16.2.6.1 | Viral Load Data – qRT-PCR/Culture |
| 16.2.6.2 | Symptom Diary Cards including Total clinical symptoms score |
| 16.2.6.3 | 24-hour tissue count & nasal discharge weight |
| 16.2.6.4 | Derived efficacy response data |
| 16.2.6.5 | Cytokine/chemokine levels |
| 16.2.6.6 | Viral resistance markers |
| 16.2.6.7 | Nasopharyngeal swab for rapid viral antigen test at discharge from quarantine |
| 16.2.6.8 | Blood - Serum ant-drug antibodies (ADA) |
| 16.2.6.9 | Community acquired virus results |
| 16.2.6.10 | HAI data |




# **Statistical Analysis Plan**

| | Safety Data |
|------------|-------------------------------------------------|
| 16.2.7 | Adverse Events |
| 16.2.7.1.1 | Solicited adverse events |
| 16.2.7.1.2 | Unsolicited Adverse Events |
| 16.2.7.1.3 | Unsolicited Serious Adverse Events |
| 16.2.7.1.4 | Unsolicited Treatment related |
| 16.2.7.1.5 | Unsolicited AE leading to study discontinuation |
| 16.2.7.1.6 | Deaths (if any) |
| 16.2.8 | Laboratory Safety Data |
| 16.2.8.1.1 | Biochemistry |
| 16.2.8.1.2 | Biochemistry – abnormal results |
| 16.2.8.2.1 | Haematology |
| 16.2.8.2.2 | Haematology – abnormal results |
| 16.2.8.3 | Urinalysis |
| 16.2.8.4 | Coagulation |
| | Other Safety Data |
| 16.2.9 | Complete and direct physical examination |
| 16.2.10 | Vital signs and tympanic temperature |
| 16.2.11 | 12-Lead Electrocardiogram |
| 16.2.12 | Spirometry |
| 16.2.13 | Reactogenicity events |

#### 13 References

- 1. Shieh G, Jan SL, and Randles RH (2006). On power and sample size determinations for the Wilcoxon–Mann–Whitney test. Journal of Nonparametric Statistics. 2006;18(1):33-43.
- 2. Hahn, G. J., & Meeker, W. Q. (2011). Statistical intervals: a guide for practitioners (Vol. 328). John Wiley & Sons.
- 3. Wilson, E. B. (1927). Probable inference, the law of succession, and statistical inference. Journal of the American Statistical Association. 22 (158): 209–212. doi:10.1080/01621459.1927.10502953


## 14 Schedule of events

| | Phase* | | | | | Inpat | ient Ph | ase (Qu | ıarantir | ie Isoli | ation ar | nd Hum | an Vira | l Challe | nge [H\ | /C]) | | | | | Outp | atient | Phase | j | ndrawal<br>it |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Screening Phase* | | Admi<br>t<br>quara | 0 | | HVC | | | Post-HVC Discharge | | | | | | | | Fo | sits | Early Withdrawal<br>Visit | | | | | | | |
| Study Day <sup>#</sup> → | Day -<br>5 | | | ing) | | | | | | D0 | | | | | | | | | | lay) | ays) | ays) | days) | days) | post<br>ge |
| Procedure <b>Ψ</b> | Day-96 to D<br>7/-6 | D-7 | D-6 | D -5 (dosing) | D-4 | D-3 | D-2 | D-1 | Pre-HVC | HVC | Post-HVC | D1 | D2 | D3 | D4 | DS | 9Q | D7 | D 8 | D17 (±1 day) | D28 (±3 days) | D60 (±7 days) | D120 (±14 days) | D180 (±14 days) | Quarantine post<br>challenge |
| Eligibility criteria (+) | Х | > | X | X <sup>(a)</sup> | | | | | | | | | | | | | | | | | | | | | |
| Written consent (b) | Х | > | X | | | | | | | | | | | | | | | | | | | | | | |
| Medical & medication history | Х | > | X | | | | | | | | | | | | | | | | | | | | | | |
| Demographics | Х | | | | | | | | | | | | | | | | | | | | | | | | |
| Height & weight, body mass index (BMI) (c) | Х | > | X | | | | | | | | | | | | | | | | (X) | | | | | (X) | (X) |
| Patient Health Questionnaire-9 (PHQ-9) | (X) | () | X) | | | | | | | | | | | | | | | | | | | | | | |
| Generalised Anxiety Disorder<br>Questionnaire-7 (GAD-7) | (X) | () | X) | | | | | | | | | | | | | | | | | | | | | | |
| Alcohol breath test | Х | > | X | | | | | | | | | | | | | | | | | | | | | | |
| Urinalysis (d) | Х | > | X | | | | | Х | | | | | | | | | | Х | | Х | Х | Χ | Х | Х | (X) |
| Urine drugs of misuse and nicotine screen | Х | > | X | | | | | | | | | | | | | | | | | | | | | | |
| Urine pregnancy test | Х | | | | | | | | | | | | | | | | | | | | Х | | | Х | (X) |
| Complete physical examination | Х | > | X | | | | | | | | | | | | | | | | Х | | | | | | (X) |
| Symptom-directed physical examination | | | | X <sup>(a)</sup> | (X) | (X) | (X) | (X) | (X) | | (X) | (X) | Х | Х | Х | (X) | (X) | (X) | | | | | | х | |




# **Statistical Analysis Plan**

| | se * | | | | | Inpat | ient Ph | ase (Qu | uarantir | ne Isola | ation ar | nd Hum | an Vira | l Challe | enge [H | VC]) | | | | | Outn | atient | Phase | | wal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pha | | | | | | | | | | | | | | | | | | | | Outp | aciciic | Tilase | | Early Withdrawal<br>Visit |
| Study Phase → | Screening Phase* | t | ission<br>o<br>antine | | Dosing with CD388 | | | | | | HVC | | | Post-HVC Discharg | | | | | | | Follow-up Clinic Visits | | | | |
| Study Day <sup>#</sup> → | ау - | | | | | | | | | D0 | | | | | | | | | | lay) | ays) | ays) | days) | days) | e post |
| Procedure <b>Ψ</b> | Day-96 to Day<br>7/-6 | D-7 | 9-Q | D -5 (dosing) | D-4 | D-3 | D-2 | D-1 | Pre-HVC | HVC | Post-HVC | D1 | D2 | D3 | D4 | DS | 90 | D7 | D 8 | D17 (±1 day) | D28 (±3 days) | D60 (±7 days) | D120 (±14 days) | D180 (±14 days) | Quarantine post<br>challenge |
| Vital signs (heart rate, respiratory rate, systolic and diastolic blood pressure, peripheral oxygen saturation [SpO <sub>2</sub> ]) (e) | Х | ) | x | X <sup>(f)</sup> | X <sup>(f)</sup> | х | х | х | х | | | х | Х | х | х | х | х | х | х | х | х | | | х | х |
| Tympanic temperature (e) | Х | > | X | X <sup>(f)</sup> | X <sup>(f)</sup> | Х | Х | 3X | | 3X | | 3X | 3X | 3X | 3X | 3X | 3X | 3X | Х | | Х | | | | Х |
| Symptom diary card (e) | | | | | | | | 3X | | 3X | | 3X | 3X | 3X | 3X | 3X | 3X | 3X | Х | | | | | | |
| 24-hour tissue count & nasal discharge weight (g) | | | | | | | | Х | Х | | | Х | Х | Х | х | Х | х | х | Х | | | | | | (X) |
| Spirometry (h) | Х | | | | | | | | | | | | | | | | | | | | | | | | |
| 12-lead electrocardiogram (ECG) | Х | ) | X | | | | | Х | | | | | | | | | | Х | | | | | | Х | (X) |
| Respiratory Tract Infection Surv | veillance | | | | | | | | | | | | | | | | | | | | | | | | |
| Weekly 7-day recall diary card (i) | | | | | | | | | | | | | | | | | | | | | | Χ | | | |
| Nasal/throat swab self-collection (j) | | | | | | | | | | | | | | | | | | | | | | (X) | | | |
| Product Administration | | | | | | | | | | | | | | | | | | | | | | | | | |
| Randomisation | X <sup>(a)</sup> | | | | | | | | | | | | | | | | | | | | | | | | |
| Investigational medicinal product (IMP; CD388/placebo) dosing | | x x | | | | | | | | | | | | | | | | | | | | | | | |
| Reactogenicity diary card (k) | x x x x x x | | | | | | | | | | | | | | | | | | | | | | | | |
| Challenge virus inoculation | | | | | | | | | | Χ | | | | | | | | | | | | | | | |
| Collection Of Blood Samples | | | | | | | | | | | | | | | | | | | | | | | | | |




# **Statistical Analysis Plan**

| | Screening Phase* | | | | | Inpat | ient Ph | ase (Qu | ıarantir | ne Isol | ation ar | nd Hum | an Vira | l Challe | nge [H\ | /C]) | | | | | Outp | atient | Phase | <u>;</u> | ıdrawal<br>t |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | ission<br>o<br>antine | | | HVC | | | | Post-HVC Discharge | | | | | | | Fe | ollow- | up Clii | nic Vis | its | Early Withdrawal<br>Visit | | | |
| Study Day # → | ау - | | | ing) | | | | | | D0 | | | | | | | | | | lay) | ays) | ays) | days) | days) | post<br>ge |
| Procedure <b>Ψ</b> | Day-96 to Day<br>7/-6 | D-7 | 9-Q | D -5 (dosing) | D-4 | D-3 | D-2 | D-1 | Pre-HVC | HVC | Post-HVC | D1 | D2 | D3 | D4 | DS | 90 | D7 | Ω | D17 (±1 day) | D28 (±3 days) | D60 (±7 days) | D120 (±14 days) | D180 (±14 days) | Quarantine post<br>challenge |
| Serum follicle-stimulating hormone (FSH) (postmenopausal women) | х | | | | | | | | | | | | | | | | | | | | | | | | |
| Serum β-human chorionic gonadotrophin (β-HCG) pregnancy test (all females) | | , | x | | | | | | | | | | | | | | | | | | | | | | |
| Human immunodeficiency virus (HIV)<br>& hepatitis serology | х | | | | | | | | | | | | | | | | | | | | | | | | |
| Haematology (I) | Х | ) | X | | | | | Х | | | | | | | | | | Х | | Х | Х | Χ | Χ | Х | (X) |
| Biochemistry (I) | Х | ) | X | | | | | Х | | | | | | | | | | Х | | Х | Χ | Χ | Χ | Х | (X) |
| Coagulation | Х | ) | X | | | | | Х | | | | | | | | | | Х | | Х | Χ | Χ | Χ | Х | (X) |
| Thyroid function test | Х | | | | | | | | | | | | | | | | | | | | | | | | |
| Cardiac enzymes | Х | | | | | | | | | | | | | | | | | | | | | | | | |
| Blood – serum markers humoral immunity (m) | Х | ) | X | | | | | | Х | | | | | | | | | | | | Х | | | | (X) |
| Blood – serum proteomics (cytokine/chemokine) (n) | | | | X <sup>(a)</sup> | | | | | Х | | | | Х | | | | | | | | | | | | |
| Blood PAXgene for transcriptomics | | | | X <sup>(a)</sup> | | | | | Х | | | | Х | Х | | | | | | | | | | | |
| Blood – plasma pharmacokinetics (PK) (n) | | | | Х | Х | | Х | | Х | | | Х | Х | Х | | | | | | Х | х | х | х | х | |
| Blood – serum anti-drug antibodies (ADA) | | | | X <sup>(a)</sup> | | | | | | | | | | | | | | | | | х | х | х | х | (X) |




# **Statistical Analysis Plan**

| | Inpatient Phase (Quarantine Isolation and Human Viral Challenge [HVC]) | | | | | | | | | | | Outpatient Phase | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Phase → | Screening Phase* | t | ission<br>o<br>antine | Dosing with CD388 | | | | | | HVC | | | Post-HVC Discharge | | | | | | | | Follow-up Clinic Visits | | | | |
| Study Day # → | Day - | | | ing) | | | | | | D0 | | | | | | | | | | lay) | ays) | ays) | days) | days) | post ge |
| Procedure <b>Ψ</b> | Day-96 to D<br>7/-6 | D-7 | 9-Q | D -5 (dosing) | D-4 | D-3 | D-2 | D-1 | Pre-HVC | HVC | Post-HVC | D1 | D2 | D3 | D4 | DS | 90 | D7 | D 8 | D17 (±1 day) | D28 (±3 days) | D60 (±7 days) | D120 (±14 days) | D180 (±14 days) | Quarantine post<br>challenge |
| Blood – PAXgene DNA for pharmacogenomics | | | | X <sup>(a)</sup> | | | | | | | | | | | | | | | | | | | | | |
| Collection Of Respiratory Samp | les | | | | | | | | | | | | | | | | | | | | | | | | |
| Nasopharyngeal swab — Respiratory<br>pathogen screen including<br>SARS-Cov-2 (e.g., Biofire) (o) | | x | | | | | | | | | | | | | | | | | | | | | | | |
| Nasopharyngeal swab – viral discharge test | | | | | | | | | | | | | | | | | | (X) | (X) | | | | | | |
| Nasopharyngeal swab for virology<br>and exploratory purposes<br>(qRT-PCR & culture, CD388) (p) | | X X X X 2X 2X 2X 2X 2X X | | | | | | | | | | | Х | Х | х | х | х | Х | (X) | | | | | | |
| Nasosorption for cytokine/chemokine (q) | | | | X <sup>(a)</sup> | | | | | Х | | | | Х | Х | | | | | | | | | | | |
| Safety Assessments | | | | | | | | | | | | | | | | | | | | | | | | | |
| Adverse event recording (r) | | | | | | | | | | | | | Cor | ntinuou | IS | | | | | | | | | | |
| Concomitant medications (r) | | Continuous | | | | | | | | | | | | | | | | | | | | | | | |



# **Statistical Analysis Plan**

#### **KEY NOTES FOR TIME AND EVENTS SCHEDULE**

| * | Results of tests or examinations performed under hVIVO generic screening process may be used to determine eligibility without the need to repeat the assessment if it is within 28 days prior to dosing with IMP. |
|---|---|
| # | With respect to challenge virus inoculation. |
| (+) | Only the applicable inclusion/exclusion criteria will be reviewed at each time point. |
| (X) | The assessment may be optional, or at the PI's discretion. The PI may perform additional safety assessments as required. |
| Х | Once, at approximately the same time each day, where applicable. |
| 2X | Twice daily, at approximately the same time each day, where applicable. |
| 3X | Three times daily, at approximately the same time each day, where applicable. |
| а | Assessments performed prior to administration of IMP. |
| b | Study-specific consent may occur on the day of admission, providing all required eligibility information has been collected through the Health Research Authority-approved hVIVO Generic Screening process. |
| С | Height will be measured at screening only. |
| d | If participant is ADA positive, additional urinalysis sample will be collected to detect haematuria and proteinuria. Additional assessments relating to ADA positive participants will be managed on a case by case basis. Participants with symptoms and signs at the respective visit may require an additional blood sample including full haematology, biochemistry, CH50 complement levels and rheumatoid factor if not already scheduled as part of the SoE. During the RTI bi-weekly call reminder, any new symptoms reported by the participant will be recorded. If a Grade 2 or higher AE is recorded, sponsor medical monitor should be notified immediately. |
| е | Apart from assessment timepoints with an (f) footnote, symptoms, temperature, and samples will be collected at approximately the same time each day (±1 hour). |
| f | On the dosing day (Day -5), vital signs and temperature will be taken 5 times: pre-dose and at 2, 6, 10 (+15 min), and 16 hours (+30 min) post-dose, and subsequently on Day -4 (24 hours [± 30min] post-dose). |
| g | Distribution of paper tissues and bags will start in the morning on Day -1 with the first collection on Day 0. Thereafter distribution and collection of tissues will occur daily, at the same time point (±1 hour) in the morning, with tissues distributed 24 hours ahead. |



| h | Eligibility only. Spirometry may be repeated at any time in the event of respiratory signs or symptoms (repeated coughing, bradypnea, tachypnoea, rales, and rhonchi) or respiratory difficulties. |
|---|---|
| i | Symptom diary cards will be completed every 7 days to capture the worst grade of symptoms that occurred over the last week. Participants will complete these from quarantine discharge until the final follow-up visit (Day 180 ±14 days), or until the resolution of a lab-confirmed influenza respiratory tract infection (RTI), whichever is first. Study site staff will contact the participants every 2 weeks to ask if an RTI has occurred and confirm that the diary cards have been completed. |
| j | Participants will be provided kits for taking nasal/throat swabs when an RTI occurs between discharge from quarantine until the final follow-up visit (Day 180 ±14 days), or until the confirmation of a lab-confirmed influenza RTI, whichever occurs first. |
| k | Collected post-dose, once daily at approximately the same time after 5 pm. |
| I | Blood will be drawn under non-fasted conditions. Repeat bloods may be drawn under fasted conditions if a lipid profile (triglyceride) or glucose is required (at the principal investigator's [PI] discretion). |
| m | Virus serology (influenza haemagglutination inhibition [HAI] assay) will be performed to determine eligibility and seroconversion. Samples may be used for related exploratory research. |
| n | Plasma PK: blood samples will be collected as outlined in Section 8.6.1. The allowable time windows for the sampling are as follows: |
| | During quarantine: |
| | O Day -5 (dosing): there is no time window requirement for the pre-dose sample |
| | O Day -5 (dosing), 2-hour time point: ±15-minute window |
| | <ul> <li>Day -5 (dosing), 4-hour time point: ±15-minute window</li> <li>Day -4 (post-dose, pre-challenge sample 1; ~24-hour time point): ±2-hour window</li> </ul> |
| | <ul> <li>Day -4 (post-dose, pre-challenge sample 1; ~24-hour time point): ±2-hour window</li> <li>Day -2 (post-dose, pre-challenge sample 2; ~72-hour time point): ±2-hour window</li> </ul> |
| | <ul> <li>Day 2 (post-dose, pre-channing sample 2, 72-hour time point): 12-hour window</li> <li>Day 0 (~120-hour time point): at approximately the same time as the viral challenge that day</li> </ul> |
| | <ul> <li>Day 1 (~144-hour time point): at approximately the same time as the first nasopharyngeal swab that day</li> </ul> |
| | <ul> <li>Day 2 (~168-hour time point): at approximately the same time as the first nasopharyngeal swab that day</li> </ul> |
| | <ul> <li>Day 3 (~192-hour time point): at approximately the same time as the first nasopharyngeal swab that day</li> </ul> |
| | After discharge from quarantine, blood PK samples will be taken at timepoints with acceptable windows as below, or until a confirmed community-acquired infection (whichever is first): |




# **Statistical Analysis Plan**

| | <ul> <li>Day 17 time point: ±1-day window</li> </ul> |
|---|---|
| | <ul> <li>Day 28 time point: ±3-day window</li> </ul> |
| | <ul> <li>Day 60 time point: ±7-day window</li> </ul> |
| | <ul> <li>Day 120 time point: ±14-day window</li> </ul> |
| | <ul> <li>Day 180 time point: ±14-day window.</li> </ul> |
| | The timepoints and number of serum proteomics sampling and PK sampling may be adjusted according to available PK data and timing of IMP relative to challenge virus inoculation. |
| 0 | Upper respiratory tract (URT) swab (e.g., nasopharyngeal swab, mid-turbinate swab, oropharyngeal swab) for respiratory virus screen to assess for the presence of other respiratory viruses; if found positive for any pathogen in the panel, the participant will not be eligible for the current quarantine. |
| p | Nasopharyngeal swabs will be taken for multiple purposes: influenza virology (PCR, and culture on those that are ≥ lower limit of quantification [LLOQ] on quantitative reverse transcriptase-polymerase chain reaction [qRT-PCR]) on Days 1 to 8 inclusive; CD388 assays on all days as per SoE. Post inoculation nasal virology samples will be collected at the same time each day during quarantine (± 1 hour). Samples may be used for related exploratory research. |
| q | Nasosorption devices will be taken for biomarkers (such as cytokines/chemokines) on all days in the morning. |
| r | Adverse events and concomitant mediations are reviewed throughout the study including pre- and post-dosing with IMP and pre- and post-influenza virus inoculation. |
| Notes: | Where any nasal sampling time points occur together, the order of sampling will typically be (1) nasosorption followed by (2) nasopharyngeal swab, with appropriate amount of time between sampling. |

| GENOMIC, TRANSCRIPTOMIC, AND PROTEOMIC SAMPLES | | | |
|---|---|---|---|
| Deoxyribonucleic acid (DNA)/ ribonucleic acid | Yes | | No |
| Deoxyribonucleic acid (DNA)/ ribonucleic acid (RNA)/ proteomic sample collection: | Nasal samples and/or blood cytokine and chemokine proteomic profile and/or mRNA profile may be assessed for associations with CD388 response, and other endpoints. Viral RNA sequencing may be performed on laboratory-confirmed positive nasal samples. | | |
| Consent considerations: | DNA pharmacogenomics may | be explored in appropriate san | nples. |




| CIDARA | CDT-CSP-001 | SAP | V2 | Final | 21 Jul 23 | docx |
|--------|-------------|-----|-----|-------|-----------|-------|
| CIDANA | CD1-C31-001 | ンヘー | v ~ | HIII | ZIJUIZJ | ·uocx |

# **Statistical Analysis Plan**

| Genetic consent. |
|---|
| Future use of remaining samples for new ethically approved health research and laboratory testing protocols according to |
| the local laws. |





## **Mock Tables and Figures**



# Cidara Therapeutics, Inc. CDT-CSP-001 / CD388.SQ.2.02

A proof-of-concept, Randomised, Double-blind, Placebo-controlled, Phase 2a Study to assess the prophylactic antiviral activity against influenza, safety, tolerability and pharmacokinetics of CD388 via a human viral challenge model

Version: v1
Date: 16DEC2022

Antoinette Anger Venn Life Sciences Biometry Services 24-26 rue de la Pépinière | 75008 Paris | France Phone: +33 1 40 21 04 10 http://www.vennlifesciences.com Antoinette.anger@vennlife.com



| <b>Document Number or Pro</b> | ect Identification: | CIDARA | CDT-CSP-003 |
|-------------------------------|---------------------|--------|-------------|

# **Mock Tables and Figures**

| ist of Tables | 3 |
|-----------------|---|
| ist of Figures4 | 2 |



Document Number or Project Identification: CIDARA\_ CDT-CSP-001

Document Version: v1

# **Mock Tables and Figures**

## List of Tables

| n° | | Enrolled | Ē | i-Eli | М | SAF | ΑI |
|---|---|---|---|---|---|---|---|
| | Demographics and Baseline characteristics | | | | | | |
| 14.1.1 | Participant disposition | Х | | | | | Х |
| 14.1.2 | Study populations and reasons for exclusion | Х | | | | | |
| 14.1.3 | Protocol deviations | | Х | | | | |
| 14.1.4.1,.2,.3,<br>.4 | Demographic data and baseline characteristics | | Х | Х | Х | Х | X (PP<br>+<br>SAF) |
| 14.1.5 | Medical History | | Х | | | | |
| 14.1.6.1,.2 | Prior Medication | | Х | | Х | | |
| 14.1.7.1,.2 | Concomitant Medication | | Х | | Х | | |
| 14.1.8.1,.2 | Compliance to Study intervention | | Х | | | Х | |
| | Efficacy | | | | | | |
| 14.2.1.1 | Primary efficacy analysis – Area under the viral load-time curve (VL-AUC) from RT-qPCR | | | | Х | | Х |
| 14.2.1.2.1, .2 | Primary efficacy, supplementary analysis – Area under the viral load-time curve (VL-AUC) from qRT-PCR | | Х | Х | | | |
| 14.2.2.1, .2 | Peak viral load from qRT-PCR | | | Х | Х | | Х |
| 14.2.3.1, .2 | Time to confirmed negative test by qRT-PCR | | | Х | Х | | Х |
| 14.2.4.1, .2 | Viral load from qRT-PCR by day and by timepoint | | Х | Х | Х | | |
| 14.2.5.1, .2 | VL-AUC from viral culture | | | Х | Х | | |
| 14.2.6.1, .2 | Peak viral load from viral culture | | | Х | Х | | |
| 14.2.7.1, .2 | Time to confirmed negative test by viral culture | | | Х | Х | | |
| 14.2.8.1, .2 | Viral load from viral culture by day and by timepoint | | Х | Х | Х | | |



| n° | | Enrolled | Ē | Ë | М | SAF | ₫ |
|---|---|---|---|---|---|---|---|
| | | Ш | | | | | |
| 14.2.9.1, .2 | Area under the curve over time of total clinical symptoms score (TSS-AUC) | | | Х | Х | | Х |
| 14.2.10.1, .2 | Peak of total clinical symptoms score (TSS) | | | Х | Х | | Х |
| 14.2.11.1, .2 | Individual peak daily total clinical symptoms score (TSS) | | | Х | Х | | |
| 14.2.12.1, .2 | Time to symptom resolution | | | Х | Х | | Х |
| 14.2.13.1,.2 | Total clinical symptoms score by day and by timepoint | | Х | Х | Х | | |
| 14.2.14.1, .2 | Incidence of confirmed influenza infection by qRT-PCR | | | Х | Х | | Х |
| 14.2.15.1, .2 | Incidence of occurrence of at least 1 positive quantitative (≥LLOQ) cell culture | | | Х | Х | | |
| 14.2.16.1, .2 | Incidence of qRT-PCR-confirmed symptomatic influenza infection | | | Х | Х | | Х |
| 14.2.17.1, .2 | Incidence of qRT-PCR-confirmed moderately severe symptomatic influenza infection | | | Х | Х | | Х |
| 14.2.18.1, .2 | Culture lab-confirmed symptomatic influenza infection | | | Х | Х | | |
| 14.2.19 | Duration of quantifiable influenza qRT-PCR measurements | | | | Х | | |
| 14.2.20 | Duration of quantifiable influenza viral culture measurements | | | | Х | | |
| 14.2.21 | Time to peak daily total clinical symptoms score | | | | Х | | |
| 14.2.22 | Total weight of mucus | | | | Х | | |
| 14.2.23 | Total number of tissues used by participants | | | | Х | | |
| 14.2.24 | Participants with symptom scored grade 2 or higher | | | | Х | | |
| 14.2.25 | Participants with symptom scored grade 2 or higher by time point | | | | Х | | |
| 14.2.26 | Participants with lab-confirmed infection and fever (≥37.9°C) | | | | Х | | |



| n° | | Enrolled | E | ITT-I | ЬР | SAF | ₹ |
|---|---|---|---|---|---|---|---|
| 14.2.27 | Laboratory-confirmed symptomatic influenza infection (community acquired) | | | | Х | | |
| 14.2.28.1 | Cytokine/chemokine levels in nasal samples | | | | Χ | | |
| 14.2.28.2 | Cytokine/chemokine levels in nasal samples (subgroup 1) | | | | Х | | |
| 14.2.28.3 | Cytokine/chemokine levels in nasal samples (subgroup 2) | | | | Х | | |
| 14.2.29.1 | Cytokine/chemokine levels in serum samples | | | | Χ | | |
| 14.2.29.2 | Cytokine/chemokine levels in serum samples (subgroup 1) | | | | Х | | |
| 14.2.29.3 | Cytokine/chemokine levels in serum samples (subgroup 2) | | | | Χ | | |
| 14.2.30 | Viral resistance markers | | | | Χ | | |
| 14.2.31.1 | Blood – Serum anti-drug antibodies (ADA) – Presence/absence of ADA | | Х | | | | |
| 14.2.31.2 | Blood – Serum anti-drug antibodies (ADA) – titer levels by day | | Х | | | | |
| | Safety | | | | | | |
| | Adverse Events | | | | | Х | |
| 14.3.1 | Summary of Adverse Events | | | | | Х | Х |
| 14.3.2.1 | Any solicited AE by SOC and PT during Period 1 | | | | | Х | |
| 14.3.2.2 | Any unsolicited TEAE by SOC and PT across all periods | | | | | Х | |
| 14.3.2.3 | Any unsolicited TEAE by SOC and PT during Period 1 | | | | | Х | |
| 14.3.2.4 | Any unsolicited TEAE by SOC and PT during Period 1 and Period 2 | | | | | Х | |
| 14.3.2.5 | Any unsolicited TEAE by SOC and PT during Period 2 | | | | | Х | |
| 14.3.2.6 | Any unsolicited TEAE by SOC and PT during Period 2 and Period 3 | | | | | Х | |
| 14.3.2.7 | Any unsolicited TEAE by SOC and PT during Period 3 | | | | | Χ | |



| n° | | Enrolled | Ē | Ė | ЬР | SAF | ΑI |
|---|---|---|---|---|---|---|---|
| 14.3.2.8 | Any unsolicited TEAE by SOC and PT during Period 3 and Period 4 | | | | | Х | |
| 14.3.3.1 | Any unsolicited TEAE across all periods by SOC, PT and relatedness | | | | | Х | Х |
| 14.3.3.2 | Any unsolicited TEAE during Period 1 by SOC, PT and relatedness | | | | | Х | |
| 14.3.3.3 | Any unsolicited TEAE during Period 1 and Period 2 by SOC, PT and relatedness | | | | | Х | |
| 14.3.3.4 | Any unsolicited TEAE during Period 2 by SOC, PT and relatedness | | | | | Х | |
| 14.3.3.5 | Any unsolicited TEAE during Period 2 and Period 3 by SOC, PT and relatedness | | | | | Х | |
| 14.3.3.6 | Any unsolicited TEAE during Period 3 by SOC, PT and relatedness | | | | | Х | |
| 14.3.3.7 | Any unsolicited TEAE during Period 3 and Period 4 by SOC, PT and relatedness | | | | | Х | |
| 14.3.4.1 | Any solicited AE by SOC/PT and maximum severity during Period 1 | | | | | Х | Х |
| 14.3.4.2 | Any unsolicited TEAE by SOC/PT and maximum severity across all periods | | | | | Х | |
| 14.3.4.3 | Any unsolicited TEAE by SOC/PT and maximum severity during Period 1 | | | | | Х | |
| 14.3.4.4 | Any unsolicited TEAE by SOC/PT and maximum severity during Period 1 and Period 2 | | | | | Х | |
| 14.3.4.5 | Any unsolicited TEAE by SOC/PT and maximum severity during Period 2 | | | | | Х | |



| n° | | Enrolled | Ē | I-III | ФФ | SAF | ΑI |
|---|---|---|---|---|---|---|---|
| 14.3.4.6 | Any unsolicited TEAE by SOC/PT and maximum severity during Period 2 and Period 3 | | | | | Х | |
| 14.3.4.7 | Any unsolicited TEAE by SOC/PT and maximum severity during Period 3 | | | | | Х | |
| 14.3.4.8 | Any unsolicited TEAE by SOC/PT and maximum severity during Period 3 and Period 4 | | | | | Х | |
| 14.3.5 | All unsolicited TEAE during Period 1 leading to study treatment discontinuation, by SOC and PT | | | | | Х | |
| 14.3.6 | Any unsolicited TEAE leading to study discontinuation, across all periods, by SOC and PT | | | | | Х | |
| 14.3.7.1 | Any unsolicited TESAE by SOC and PT across all periods | | | | | Χ | |
| 14.3.7.2 | Any SAE by SOC and PT during Period 1 | | | | | Χ | |
| 14.3.7.3 | Any SAE by SOC and PT during Period 1 and Period 2 | | | | | Х | |
| 14.3.7.4 | Any SAE by SOC and PT during Period 2 | | | | | Χ | |
| 14.3.7.5 | Any SAE by SOC and PT during Period 2 and Period 3 | | | | | Х | |
| 14.3.7.6 | Any SAE by SOC and PT during Period 3 | | | | | Х | |
| 14.3.7.7 | Any SAE by SOC and PT during Period 3 and Period 4 | | | | | Х | |
| 14.3.8 | Any SAE by SOC, PT and relatedness across all periods | | | | | Х | |
| | Laboratory Safety | | | | | Χ | |
| 14.3.9.1.1 | Laboratory Safety: quantitative descriptive statistics | | | | | Х | |
| 14.3.9.1.2 | Laboratory Safety: quantitative descriptive statistics – Change from baseline | | | | | Х | |
| 14.3.9.2 | Laboratory Safety: Shift tables | | | | | Х | |
| 14.3.9.3 | Laboratory Safety: Subjects with at least a 2-grade increase from baseline at any post-baseline | | | | | Х | |



Document Number or Project Identification: CIDARA\_ CDT-CSP-001


| n° | | Enrolled | E | H | dd | SAF | Ā |
|---|---|---|---|---|---|---|---|
| 14.3.9.4 | Laboratory Safety: Urinalysis | | | | | X | |
| | Vital Signs and Tympanic Temperature | | | | | Х | |
| 14.3.10.1 | Vital Signs and Tympanic Temperature: quantitative descriptive statistics | | | | | Х | |
| 14.3.10.2 | Vital Signs and Tympanic Temperature: quantitative descriptive statistics – Change from baseline | | | | | Х | |
| 14.3.10.3 | Vital Signs and Tympanic Temperature: qualitative descriptive statistics | | | | | Х | |
| | 12-Lead Electrocardiogram | | | | | Х | |
| 14.3.11.1.1 | 12-Lead ECG: quantitative descriptive statistics | | | | | Х | |
| 14.3.11.1.2 | 12-Lead ECG: quantitative descriptive statistics – change from baseline | | | | | Х | |
| 14.3.11.2 | 12-Lead ECG: qualitative descriptive statistics | | | | | Х | |



Document Number or Project Identification: CIDARA\_ CDT-CSP-001


# **Mock Tables and Figures**

n / N

#### Table 14.1.1: Participant Disposition

#### Enrolled Analysis Set

| Description | Statistics | PLACEBO<br>(N=XX) | CD388 XX MG<br>(N=XX) | CD388 150 MG<br>(N=XX) | All<br>(N=XX) |
|---|---|---|---|---|---|
| Randomized participants | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Participants receiving treatment | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Participants receiving challenge virus | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Participants who completed the study | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes<br>No | n (%)<br>n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| If discontinued, reason for study discontinuation | И | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| Death | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Adverse event or Serious adverse event | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Withdrawal by subject | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Investigator's decision | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Non-compliance with study requirements | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Pregnancy | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Study terminated by Sponsor | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to follow-up | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Study duration (days) | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | S.D | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |



| <b>Document Number</b> | or Project | Identification: | $CID\Delta R\Delta$ | CDT-CSP-00 |
|---|---|---|---|---|
| Document Number | or Froject | iuentincation. | CIDANA | CD1-C3F-00. |

# **Mock Tables and Figures**

n / N

#### Table 14.1.1: Participant Disposition

#### Enrolled Analysis Set

| Dogarintion | 0++++++ | PLACEBO | CD388 XX MG | CD388 150 MG | All |
|-------------|------------|---------|-------------|--------------|--------|
| Description | Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) |

S.D = Standard Deviation - Q1 = First Quartile - Q3 = Third Quartile Percentages are based on the number of subjects without missing values in the Enrolled analysis set

Data source(s): addmain.xxxx (Date time)
Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)
Program: /Study/tlf/tf/pgm/pgm\_name.sas Date time / run Date time by Stat\_name


Document Number or Project Identification: CIDARA\_CDT-CSP-001


# **Mock Tables and Figures**

n / N

### Table 14.1.2: Study Populations and Reasons for Exclusion

#### Enrolled Analysis Set

| Description | Statistics | PLACEBO<br>(N=XX) | CD388 XX MG<br>(N=XX) | CD388 150 MG<br>(N=XX) | All<br>(N=XX) |
|---|---|---|---|---|---|
| | | (N-AA) | (N-AA) | (N-AA) | (IV-AA) |
| Enrolled | N | XX | XX | XX | XX |
| Intent-To-Treat (ITT) | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| Yes | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason for exclusion from ITT | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| Not Randomized | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not study treatment administered | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Intent-To-Treat Infected (ITT-I) | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| Yes | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason for exclusion from ITT-I | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| Not Randomized | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not study treatment administered | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| - | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Per-Protocol (PP) | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| Yes | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason for exclusion from PP | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| Not Randomized | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not study treatment administered | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |




Document Number or Project Identification: CIDARA\_ CDT-CSP-001


## **Mock Tables and Figures**

n / N

#### Table 14.1.2: Study Populations and Reasons for Exclusion

#### Enrolled Analysis Set

| Description | Statistics | | JACEBO<br>N=XX) | | 88 XX MG<br>N=XX) | | 8 150 MG<br>N=XX) | ( | All<br>N=XX) |
|---|---|---|---|---|---|---|---|---|---|
| Not challenge inoculated | n (%) | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Not have a valid result at least 80% of the planned gRT-PCR nasal samples | ofn (%) | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| At least one major protocol deviation likely to impact the evaluation the primary endpoint | n (%)<br>on | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Safety Analysis Set (SAF) | N | | XX | | XX | | XX | | XX |
| | Missing | | XX | | XX | | XX | | XX |
| Yes | n (%) | | (XX.X) | | (XX.X) | XX | (XX.X) | | (XX.X) |
| No | n (%) | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Reason for exclusion from SAF | N | | XX | | XX | | XX | | XX |
| | Missing | | XX | | XX | | XX | | XX |
| Not study treatment administrated | n (%) | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |

Percentages are based on the number of subjects without missing values in the Enrolled analysis set except for reason for exclusion where the percentages are based on subjects not included without missing values in the corresponding population

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time) Program: /Study/tlf/tf/pgm/pgm\_name.sas Date time / run Date time by Stat\_name




Document Number or Project Identification: CIDARA\_ CDT-CSP-001


# **Mock Tables and Figures**

n / N

#### Table 14.1.3: Protocol Deviations

#### ITT Analysis Set

| Minan an Maian | PLACEBO | CD388 XX MG | CD388 150 MG | All |
|---|---|---|---|---|
| Minor or Major | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Deviation Category | n (%) [d] | n (%) [d] | n (%) [d] | n (%) [d] |
| Any protocol deviation | xx (xx.x) [xx] | xx (xx.x) [xx] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Major protocol deviation | xx (xx.x) [xx] | xx (xx.x) [xx] | xx (xx.x) [xx] | XX (XX.X) [XX] |
| Major deviation 1 | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Major deviation 2 | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Major deviation n | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Minor protocol deviation | xx (xx.x) [xx] | xx (xx.x) [xx] | xx (xx.x) [xx] | XX (XX.X) [XX] |
| Minor deviation 1 | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Minor deviation 2 | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Minor deviation n | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |

d = number of deviations

Percentages are based on the number of subjects in the Intent to Treat (ITT) analysis set

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time) Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name


# **Mock Tables and Figures**

n / N

Table 14.1.4.1: Demographics and Baseline Characteristics

## ITT Analysis Set

| Description | Statistics | PLACEBO | CD388 XX MG | CD388 150 MG | All |
|---|---|---|---|---|---|
| | | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Sex | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| Male | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Female | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Age | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | S.D | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Ethnicity | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| Hispanic / Latino | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Hispanic / Latino | n (응) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Race | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| Asian | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Black or African American | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| White | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Hawaiian or Pacific Islander | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Native Indian or Alaskan | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | n (% | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Weight (kg) | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |


# **Mock Tables and Figures**

n / N

### Table 14.1.4.1: Demographics and Baseline Characteristics

## ITT Analysis Set

| Description | Statistics | PLACEBO | CD388 XX MG | CD388 150 MG | All |
|---|---|---|---|---|---|
| 1 | | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| | S.D | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Height (cm) | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | S.D | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| BMI (kg/m²) | N | XX | XX | XX | XX |
| , 3, , | Missing | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | S.D | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX |
| | Min, Max | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |

S.D = Standard Deviation - Q1 = First Quartile - Q3 = Third Quartile

Percentages are based on the number of subjects without missing values in the Intent to Treat (ITT) Analysis Set

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)

Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name

### This mock table is used for the following tables:





# **Mock Tables and Figures**

Table 14.1.4.2: Demographics and Baseline Characteristics - ITT-I Analysis Set Table 14.1.4.3: Demographics and Baseline Characteristics - PP Analysis Set Table 14.1.4.4: Demographics and Baseline Characteristics - SAF Analysis Set





# **Mock Tables and Figures**

n / N

## Table 1.4.5: Medical History

## ITT Analysis Set

| | PLACEBO | CD388 XX MG | CD388 150 MG | All |
|---|---|---|---|---|
| System Organ Class Preferred Term | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Preferred Term | n (%) | n (%) | n (%) | n (%) |
| any Medical History | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| OC A | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PT a | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PT b | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| SOC B | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PT c | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PT d | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Percentages are based on the number of subjects in the Intent to Treat (ITT) Analysis Set
Subjects with the same System Organ Class and Preferred Term will be counted only once within the SOC and PT
Coding dictionnary: MedDRA version xx.x (Month year)

Data source(s): addmain.xxxx (Date time)
Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)

Program: /Study/tlf/tf/pgm/pgm\_name.sas Date time / run Date time by Stat\_name


## **Mock Tables and Figures**

n / N

#### Table 1.4.6.1: Prior Medication

#### ITT Analysis Set

| .mc .t1 2 | PLACEBO | CD388 XX MG | CD388 150 MG | All |
|----------------------|-----------|-------------|--------------|-----------|
| ATC Level 2 | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Preferred Name | n (%) | n (%) | n (%) | n (%) |
| any Prior Medication | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ATC Level 2 A | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PN a | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PN b | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ATC Level 2 B | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PN C | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| PN d | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Percentages are based on the number of subjects in the Intent to Treat (ITT) Analysis Set Subjects with the same Anatomical Term Class and Preferred Name will be counted only once within the ATC and PN Coding Dictionary: WHODrug Global version (Month day, year)

Data source(s): addmain.xxxx (Date time)
Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)
Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name

### This mock table is used for the following tables:

Table 14.1.6.2: Concomitant Medications - PP Analysis Set Table 14.1.7.1: Concomitant Medications - ITT Analysis Set Table 14.1.7.2: Concomitant Medications - PP Analysis Set




| Document Number or Pro | ject Identification: | CIDARA | CDT-CSP- | 001 |
|------------------------|----------------------|--------|----------|-----|

# **Mock Tables and Figures**

n / N

### Table 14.1.8.1: Compliance to Study Intervention

## ITT Analysis Set

| Ctatiotics | PLACEBO | CD388 XX MG | CD388 150 MG | All |
|---|---|---|---|---|
| Statistics (N=XX) | | (N=XX) | (N=XX) | (N=XX) |
| N | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX |
| n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | n (%) | N XX Missing XX n (%) XX (XX.X) | N XX XX Missing XX XX n (%) XX (XX.X) XX (XX.X) | N XX XX XX XX Missing XX XX XX XX n (%) XX (XX.X) XX (XX.X) XX (XX.X) |

Percentages are based on the number of subjects without missing values in the Intent-To-Treat (ITT) Analysis Set

Data source(s): addmain.xxxx (Date time)
Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)

Program: /Study/tlf/tf/pgm/pgm\_name.sas Date time / run Date time by Stat\_name

## Table 14.1.8.2: Compliance to Study Intervention - SAF Analysis Set





## **Mock Tables and Figures**

n / N

Table 14.2.1.1: Primary efficacy - Area Under the Viral Load-time Curve (VL-AUC) from qRT-PCR

PP Analysis Set

| Description | Statistics | PLACEBO | CD388 XX MG | CD388 150 MG | ALL |
|---|---|---|---|---|---|
| Description | Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Area under the viral load-time | N | XX | XX | XX | XX |
| curve (VL-AUC) from qRT-PCR | Missing | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | S.D | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | 95% CI Mean | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] |
| CD388 doses vs. Placebo comparison | Hodges-Lehmann estimation of the location shift | | XX.X | xx.x | |
| - | (95% CI) | | [XX.X; XX.X] | [XX.X; XX.X] | |
| | P-value for one-sided Wilcoxon rank sum test | | X.XXXX | X.XXXX | |

S.D = Standard Deviation - Q1 = First Quartile - Q3 = Third Quartile - CI = Confidence Interval

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)
Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name

### This mock table is used for the following tables:

Table 14.2.1.2.1: Primary efficacy, supplementary analysis - Area Under the Viral Load-time Curve (VL-AUC) from qRT-PCR- ITT Analysis Set

Table 14.2.1.2.2: Primary efficacy, supplementary analysis - Area Under the Viral Load-time Curve (VL-AUC) from qRT-PCR-ITT-I Analysis Set

Table 14.2.5.1: Area Under the Viral Load-time Curve (VL-AUC) from Viral Culture - PP Analysis Set




# **Mock Tables and Figures**

Table 14.2.5.2: Area Under the Viral Load-time Curve (VL-AUC) from Viral Culture - ITT-I Analysis Set





## **Mock Tables and Figures**

n / N

### Table 14.2.2.1: Peak Viral Load from qRT-PCR

## PP Analysis Set

| Obabiatia. | PLACEBO | CD388 XX MG | CD388 150 MG | ALL |
|---|---|---|---|---|
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| N | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| S.D | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| 95% CI Mean | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] |
| Difference in means vs. Placebo | | XX.XX | XX.XX | |
| 95% CI | | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | |
| P-value for one-sided Wilcoxon rank sum test | | X.XXX | X.XXXX | |
| | Missing Mean S.D Median Q1, Q3 Min, Max 95% CI Mean Difference in means vs. Placebo | N XX Missing XX Mean XX.XX S.D XX.XX Median XX.XX Median XX.XX Min, Max XX.X, XX.X Difference in means vs. Placebo 95% CI P-value for one-sided Wilcoxon | N XX XX Missing XX XX Mean XX.XX XX.XX S.D XX.XX XX.XX Median XX.XX XX.XX Q1, Q3 XX.X, XX.X XX.X, XX.X Min, Max XX.X, XX.X XX.X, XX.X 95% CI Mean [XX.XX; XX.XX] [XX.XX; XX.XX] Difference in means vs. Placebo XX.XX 95% CI [XX.XX; XX.XX] P-value for one-sided Wilcoxon X.XXXX | Statistics (N=XX) (N=XX) (N=XX) N XX XX XX Missing XX XX XX XX Mean XX.XX XX.XX XX.XX XX.XX S.D XX.XX XX.XX XX.XX XX.XX Median XX.XX XX.XX XX.XX XX.XX Q1, Q3 XX.XX, XX.X XX.XX, XX.X XX.XX XX.XX XX.XX Min, Max XX.XX, XX.X XX.XX XX.XXX XX.XXXX XX.XXXX XX.XXXX XX.XXX |

S.D = Standard Deviation - Q1 = First Quartile - Q3 = Third Quartile - CI = Confidence Interval

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)
Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name

### This mock table is used for the following tables:

Table 14.2.2.2: Peak Viral Load from qRT-PCR - ITT-I Analysis Set

Table 14.2.6.1: Peak Viral Load from Viral Culture- PP Analysis Set

Table 14.2.6.2: Peak Viral Load from Viral Culture - ITT-I Analysis Set





# **Mock Tables and Figures**

Table 14.2.9.1: Area Under the Curve over time of Total Clinical Symptoms Score (TSS-AUC) - PP Analysis Set Table 14.2.9.2: Area Under the Curve over time of Total Clinical Symptoms Score (TSS-AUC) - ITT-I Analysis Set Table 14.2.10.1: Peak of Total Clinical Symptoms Score (TSS) - PP Analysis Set Table 14.2.10.2: Peak of Total Clinical Symptoms Score (TSS) - ITT-I Analysis Set Table 14.2.11.1: Individual Peak Daily Total Clinical Symptoms Score (TSS) - PP Analysis Set Table 14.2.11.2: Individual Peak Daily Total Clinical Symptoms Score (TSS) - ITT-I Analysis Set


# **Mock Tables and Figures**

n / N

Table 14.2.3.1: Time to Confirmed Negative Test by qRT-PCR

PP Analysis Set

| Description | Statistics | PLACEBO<br>(N=XX) | CD388 XX MG<br>(N=XX) | CD388 150 MG<br>(N=XX) |
|---|---|---|---|---|
| Number of subjects | | | | |
| With event | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Censored | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Number of subjects who do not<br>have a detectable qRT-PCR<br>value | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Kaplan-Meier Estimates of | 25th Percentile (95% CI) | XX [XX ; XX] | XX [XX ; XX] | XX [XX ; XX] |
| Time to confirmed negative | Median (95% CI) | XX [XX ; XX] | XX [XX ; XX] | XX [XX ; XX] |
| test by qRT-PCR (hours) | 75th Percentile (95% CI) | XX [XX ; XX] | XX [XX ; XX] | XX [XX ; XX] |
| Kaplan-Meier estimates (%) | 0 hour | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) |
| (95% CI) of the cumulative | 12 hours | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) |
| proportion of subjects with | 24 hours | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) |
| an event: | 36 hours | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) |
| | 48 hours | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) | XX.X (XX.X; XX.X) |
| | P-value for one-sided Gehan-Wilcoxon test | | X.XXXX | X.XXXX |

CI = Confidence Interval

Percentages are based on the number of subjects in the Per Protocol (PP) Analysis Set

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time) Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name





## **Mock Tables and Figures**

## This mock table is used for the following tables:

Table 14.2.3.2: Time to Confirmed Negative Test by qRT-PCR - ITT-I Analysis Set

Table 14.2.7.1: Time to Confirmed Negative Test by Viral Culture - PP Analysis Set

Table 14.2.7.2: Time to Confirmed Negative Test by Viral Culture - ITT-I Analysis Set

Table 14.2.12.1: Time to Symptom Resolution - PP Analysis Set

Table 14.2.12.2: Time to Symptom Resolution - ITT-I Analysis Set


## **Mock Tables and Figures**

n / N

Table 14.2.4.1: Viral Load from qRT-PCR by day and by timepoint

#### PP Analysis Set

| Description | Statistics | PLACEBO | CD388 XX MG | CD388 150 MG | All |
|---|---|---|---|---|---|
| | | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| sit X* | N | XX | XX | XX | XX |
| 510 11 | Missing | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | S.D | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| sit X* | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | S.D | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

S.D = Standard Deviation - Q1 = First Quartile - Q3 = Third Quartile

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time) Program:  $Study/tlf/tf/pgm/pgm_name.sas$  Date time / run Date time by  $Stat_name$ 

Note: \* Visit X can be "Day X - Timepoint X" or "Day X"

### This mock table is used for the following tables:

Table 14.2.4.2: Viral Load from qRT-PCR by day and by timepoint - ITT Analysis Set Table 14.2.4.3: Viral Load from qRT-PCR by day and by timepoint - ITT-I Analysis Set





# **Mock Tables and Figures**

```
Table 14.2.8.1: Viral Load from Viral Culture by day and by timepoint - PP Analysis Set
Table 14.2.8.2: Viral Load from Viral Culture by day and by timepoint - ITT Analysis Set
Table 14.2.8.3: Viral Load from Viral Culture by day and by timepoint - ITT-I Analysis Set
Table 14.2.13.1: Total Clinical Symptoms Score by day and by timepoint - PP Analysis Set
Table 14.2.13.2: Total Clinical Symptoms Score by day and by timepoint - ITT Analysis Set
Table 14.2.13.3: Total Clinical Symptoms Score by day and by timepoint - ITT-I Analysis Set
Table 14.2.28.1: Cytokine/Chemokine Levels in Nasal Samples - PP Analysis Set
Table 14.2.28.2: Cytokine/Chemokine Levels in Nasal Samples (subgroup 1) - PP Analysis Set
Table 14.2.28.3: Cytokine/Chemokine Levels in Nasal Samples (subgroup 2) - PP Analysis Set
Table 14.2.29.1: Cytokine/Chemokine Levels in Serum Samples - PP Analysis Set
Table 14.2.29.2: Cytokine/Chemokine Levels in Serum Samples (subgroup 1) - PP Analysis Set
Table 14.2.29.3: Cytokine/Chemokine Levels in Serum Samples (subgroup 2) - PP Analysis Set
Table 14.2.31.2: Blood - Serum Anti-drug Antibodies (ADA) - Titer Levels by day - ITT Analysis Set
Table 14.3.9.1.1: Laboratory Safety: quantitative descriptive statistics - SAF Analysis Set
Table 14.3.9.1.2: Laboratory Safety: quantitative descriptive statistics - Change from Baseline - SAF Analysis Set
Table 14.3.9.4: Laboratory Safety: Urinalysis: quantitative descriptive statistics - SAF Analysis Set
Table 14.3.10.1: Vital Signs and Tympanic Temperature: quantitative descriptive statistics - SAF Analysis Set
Table 14.3.10.2: Vital Signs and Tympanic Temperature: quantitative descriptive statistics - Change from Baseline -
SAF Analysis Set
Table 14.3.11.1: 12-Lead ECG: quantitative descriptive statistics - SAF Analysis Set
Table 14.3.11.1.2: 12-Lead ECG: quantitative descriptive statistics - Change from Baseline - SAF Analysis Set
```


## **Mock Tables and Figures**

n / N

Table 14.2.14.1: Incidence of Confirmed Influenza Infection by qRT-PCR

### PP Analysis Set

| Description | Statistics | PLACEBO<br>(N=XX) | CD388 XX MG<br>(N=XX) | CD388 150 MG<br>(N=XX) | All<br>(N=XX) |
|---|---|---|---|---|---|
| qRT-PCR-confirmed influenza | N | XX | XX | XX | XX |
| infection | Missing | XX | XX | XX | XX |
| No | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 95% CI | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] |
| Yes | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 95% CI | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] |
| CD388 doses vs. Placebo comparison | One-sided Fisher's exact p-value | | x.xxxx | x.xxxx | |

CI = Confidence Interval

Percentages are based on the number of subjects without missing values in the Per Protocol (PP) Analysis Set

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time) Program:  $/Study/tlf/tf/pgm/pgm_name.sas$  Date time / run Date time by  $Stat_name$ 

### This mock table is used for the following tables:

Table 14.2.14.2: Incidence of Confirmed Influenza Infection by qRT-PCR - ITT-I Analysis Set

Table 14.2.15.1: Incidence of Occurrence of At Least 1 Positive Quantitative (≥LLOQ) Cell Culture - PP Analysis Set

Table 14.2.15.2: Incidence of Occurrence of At Least 1 Positive Quantitative (≥LLOQ) Cell Culture - ITT-I Analysis

Set

Table 14.2.16.1: Incidence of qRT-PCR-Confirmed Symptomatic Influenza Infection - PP Analysis Set

Table 14.2.16.2: Incidence of qRT-PCR-Confirmed Symptomatic Influenza Infection - ITT-I Analysis Set





# **Mock Tables and Figures**

Table 14.2.17.1: Incidence of qRT-PCR-Confirmed Moderately Severe Symptomatic Influenza Infection - PP Analysis Set Table 14.2.17.2: Incidence of qRT-PCR-Confirmed Moderately Severe Symptomatic Influenza Infection - ITT-I Analysis Set Table 14.2.18.1: Incidence of Culture Lab-Confirmed Symptomatic Influenza Infection - PP Analysis Set Table 14.2.18.2: Incidence of Culture Lab-Confirmed Symptomatic Influenza Infection - ITT-I Analysis Set





## **Mock Tables and Figures**

n / N

## Table 14.2.19: Duration of Quantifiable Influenza qRT-PCR Measurements

#### PP Analysis Set

| Description | Statistics | PLACEBO<br>(N=XX) | CD388 XX MG<br>(N=XX) | CD388 150 MG<br>(N=XX) | All<br>(N=XX) |
|---|---|---|---|---|---|
| | | (14 1111) | (14 1111) | (14 1111) | (14 2121) |
| ration of quantifiable influenza | N | XX | XX | XX | XX |
| T-PCR measurements (hours) | Missing | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | S.D | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | 95% CI Mean | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX |

S.D = Standard Deviation - Q1 = First Quartile - Q3 = Third Quartile - CI = Confidence Interval

Data source(s): addmain.xxxx (Date time)

#### This mock table is used for the following tables:

Table 14.2.20: Duration of Quantifiable Influenza Viral Culture Measurements - PP Analysis Set

Table 14.2.21: Time to Peak Daily Total Clinical Symptoms Score - PP Analysis Set

Table 14.2.22: Total Weight of Mucus - PP Analysis Set

Table 14.2.23: Total Number of Tissues Used by Participants - PP Analysis Set





## **Mock Tables and Figures**

n / N

## Table 14.2.24: Participants with Symptom Scored Grade 2 or higher

#### PP Analysis Set

| Description | Statistics | PLACEBO<br>(N=XX) | CD388 XX MG<br>(N=XX) | CD388 150 MG<br>(N=XX) | All<br>(N=XX) |
|---|---|---|---|---|---|
| Participants with symptom | N | XX | XX | XX | XX |
| scored grade 2 or higher | Missing | XX | XX | XX | XX |
| No | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 95% CI | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] |
| Yes | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 95% CI | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] | [XX.XX ; XX.XX] |

CI = Confidence Interval

Percentages are based on the number of subjects without missing values in the Per Protocol (PP) Analysis Set

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time) Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name

#### This mock table is used for the following tables:

Table 14.2.26: Participants with Lab-Confirmed Infection and Fever (≥37.9°C) - PP Analysis Set

Table 14.2.27: Laboratory-Confirmed Symptomatic Influenza Infection (community acquired) - PP Analysis Set





## **Mock Tables and Figures**

n / N

Table 14.2.25: Participants with Symptom Scored Grade 2 or higher by day

#### PP Analysis Set

| Description | Statistics | PLACEBO<br>(N=XX) | CD388 XX MG<br>(N=XX) | CD388 150 MG<br>(N=XX) | All<br>(N=XX) |
|---|---|---|---|---|---|
| | (IV-VV) | (IV-AA) | (N-VV) | (IN-XX) | |
| isit X | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| No** | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes** | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| isit X | N | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| No** | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes** | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Percentages are based on the number of subjects without missing values in the Per Protocol (PP) Analysis Set

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)

Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name

Note: \* Visit X can be "Day X - Timepoint X" or "Day X"

Note: \*\* Modalities updated according to analysis

#### This mock table is used for the following tables:

Table 14.2.30: Viral Resistance Markers - PP Analysis Set

Table 14.2.31.1: Blood - Serum Anti-Drug Antibodies (ADA) - Titer Levels by day - ITT Analysis Set

Table 14.3.9.2: Laboratory Safety: Shift tables - SAF Analysis Set

Table 14.3.9.3: Laboratory Safety: Subjects with at least a 2-grade increase from baseline at any post-baseline - SAF Analysis Set

Table 14.3.9.4: Laboratory Safety: Urinalysis: qualitative descriptive statistics - SAF Analysis Set




| <b>Document Number or Pro</b> | ect Identification: | CIDARA | CDT-CSP-003 |
|-------------------------------|---------------------|--------|-------------|

# **Mock Tables and Figures**

Table 14.3.10.3: Vital Signs and Tympanic Temperature: qualitative descriptive statistics - SAF Analysis Set Table 14.3.11.2: 12-Lead ECG: qualitative descriptive statistics - SAF Analysis Set


# **Mock Tables and Figures**

n / N

## Table 14.3.1: Summary of Adverse Events

## SAF Analysis Set

| Description | PLACEBO<br>(N=XX)<br>n (%) [e] | CD388 XX MG<br>(N=XX)<br>n (%) [e] | CD388 150 MG<br>(N=XX)<br>n (%) [e] | ALL<br>(N=XX)<br>n (%) [e] |
|---|---|---|---|---|
| Any AE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Period 1: | | | | |
| Any TEAE (solicited and unsolicited) | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any solicited AE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE - leading to study treatment discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE leading to study discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE considered as related to study treatment (at least possibly related) | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any SAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Period 1 and Period 2: | | | | |
| Any unsolicited TEAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE leading to study discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE considered as related to study treatment (at least possibly related) | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any SAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |


# **Mock Tables and Figures**

n / N

## Table 14.3.1: Summary of Adverse Events

## SAF Analysis Set

| Description | PLACEBO<br>(N=XX)<br>n (%) [e] | CD388 XX MG<br>(N=XX)<br>n (%) [e] | CD388 150 MG<br>(N=XX)<br>n (%) [e] | ALL<br>(N=XX)<br>n (%) [e] |
|---|---|---|---|---|
| Period 2: | | | | |
| Any unsolicited TEAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE leading to study discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE considered as related to study treatment (at least possibly related) | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any SAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Period 2 and Period 3: | | | | |
| Any unsolicited TEAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE leading to study discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE considered as related to study treatment (at least possibly related) | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any SAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Period 3: | | | | |
| Any unsolicited TEAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE leading to study discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE considered as related to study treatment (at least possibly related) | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |


# **Mock Tables and Figures**

n / N

## Table 14.3.1: Summary of Adverse Events

## SAF Analysis Set

| Description | PLACEBO<br>(N=XX)<br>n (%) [e] | CD388 XX MG<br>(N=XX)<br>n (%) [e] | CD388 150 MG<br>(N=XX)<br>n (%) [e] | ALL<br>(N=XX)<br>n (%) [e] |
|---|---|---|---|---|
| Any SAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Period 3 and Period 4: | | | | |
| Any unsolicited TEAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE leading to study discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE considered as related to study treatment (at least possibly related) | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any SAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Period 4 | | | | |
| Any unsolicited TEAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE leading to study discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE considered as related to study treatment (at least possibly related) | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any SAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Across all Periods: | | | | |
| Any unsolicited TEAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any unsolicited TEAE leading to study discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |





# **Mock Tables and Figures**

n / N

### Table 14.3.1: Summary of Adverse Events

## SAF Analysis Set

| | PLACEBO | CD388 XX MG | CD388 150 MG | ALL |
|---|---|---|---|---|
| Description | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| | n (%) [e] | n (%) [e] | n (%) [e] | n (%) [e] |
| Any unsolicited TEAE considered as related to study treatment (at least possibly related) | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any SAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any TESAE leading to study treatment permanent discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any TESAE leading to study discontinuation | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Any TESAE considered related to the study treatment | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Death | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |

e = number of events

Percentages are based on the number of subjects in the Safety (SAF) Analysis Set Presented: number of subjects (percent of subjects) [number of events]

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time) Program:  $/Study/tlf/tf/pgm/pgm_name.sas$  Date time / run Date time by  $Stat_name$ 





## **Mock Tables and Figures**

n / N

#### Table 14.3.2.1: Any Solicited AE by SOC and PT during Period 1

#### SAF Analysis Set

| 2 | PLACEBO | CD388 XX MG | CD388 150 MG | All |
|---|---|---|---|---|
| System Organ Class | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Preferred Term | n (%) [e] | n (%) [e] | n (%) [e] | n (%) [e] |
| Any solicited AE | xx (xx.x) [xx] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| SOC A | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | xx (xx.x) [xx] |
| PT a | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| PT b | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| SOC B | XX (XX.X) [XX] | xx (xx.x) [xx] | xx (xx.x) [xx] | xx (xx.x) [xx] |
| PT c | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| PT d | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |

e = number of events

Percentages are based on the number of subjects in the Safety (SAF) Analysis Set Subjects with the same System Organ Class and Preferred Term will be counted only once within the SOC and PT Coding dictionnary: MedDRA version xx.x (Month year)

Data source(s): addmain.xxxx (Date time)
Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)
Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name

### This mock table is used for the following tables:

Table 14.3.2.2: Any Unsolicited TEAE by SOC and PT across all Periods - SAF Analysis Set Table 14.3.2.3: Any Unsolicited TEAE by SOC and PT during Period 1 - SAF Analysis Set

Table 14.3.2.4: Any Unsolicited TEAE by SOC and PT during Period 1 and Period 2 - SAF Analysis Set

Document Template: SOP-CORP-01 AP02 V01





# **Mock Tables and Figures**

```
Table 14.3.2.5: Any Unsolicited TEAE by SOC and PT during Period 2 - SAF Analysis Set
Table 14.3.2.6: Any Unsolicited TEAE by SOC and PT during Period 2 and Period 3 - SAF Analysis Set
Table 14.3.2.7: Any Unsolicited TEAE by SOC and PT during Period 3 - SAF Analysis Set
Table 14.3.2.8: Any Unsolicited TEAE by SOC and PT during Period 3 and Period 4 - SAF Analysis Set
Table 14.3.5: All Unsolicited TEAE during Period 1 Leading to Study Treatment Discontinuation, by SOC and PT - SAF
Analysis Set
Table 14.3.6: Any Unsolicited TEAE Leading to Study Discontinuation, across all Periods, by SOC and PT - SAF
Analysis Set
Table 14.3.7.1: Any Unsolicited TESAE by SOC and PT across all Periods - SAF Analysis Set
Table 14.3.7.2: Any SAE by SOC and PT during Period 1 - SAF Analysis Set
Table 14.3.7.3: Any SAE by SOC and PT during Period 2 - SAF Analysis Set
Table 14.3.7.4: Any SAE by SOC and PT during Period 2 - SAF Analysis Set
Table 14.3.7.5: Any SAE by SOC and PT during Period 2 - SAF Analysis Set
Table 14.3.7.6: Any SAE by SOC and PT during Period 3 - SAF Analysis Set
Table 14.3.7.6: Any SAE by SOC and PT during Period 3 - SAF Analysis Set
Table 14.3.7.7: Any SAE by SOC and PT during Period 3 - SAF Analysis Set
```





# **Mock Tables and Figures**

n / N

Table 14.3.3.1: Any Unsolicited TEAE across all Periods by SOC, PT and Relatedness

SAF Analysis Set

| System Organ Class | PLACEBO | CD388 XX MG | CD388 150 MG | ALL |
|---|---|---|---|---|
| Preferred Term | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Relatedness | n (%) [e] | n (%) [e] | n (%) [e] | n (%) [e] |
| Any unsolicited TEAE | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Unrelated | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Related | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| SOC A | XX (XX.X) [XX] | xx (xx.x) [xx] | XX (XX.X) [XX] | xx (xx.x) [xx] |
| PT a | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Unrelated | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Related | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| PT b | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Unrelated | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Related | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| SOC B | XX (XX.X) [XX] | xx (xx.x) [xx] | XX (XX.X) [XX] | xx (xx.x) [xx] |
| PT c | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Unrelated | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Related | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| PT d | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Unrelated | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |
| Related | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] | XX (XX.X) [XX] |

•••



| <b>Document Number or Pro</b> | ject Identification: | CIDARA | CDT-CSP-00 |
|---|---|---|---|
|---|---|---|---|

# **Mock Tables and Figures**

n / N

Table 14.3.3.1: Any Unsolicited TEAE across all Periods by SOC, PT and Relatedness

### SAF Analysis Set

| System Organ Class | PLACEBO | CD388 XX MG | CD388 150 MG | ALL |
|--------------------|-----------|-------------|--------------|-----------|
| Preferred Term | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Relatedness | n (%) [e] | n (%) [e] | n (%) [e] | n (%) [e] |

e = number of events

Percentages are based on the number of subjects in the Safety (SAF) Analysis Set

Subjects with the same System Organ Class and Preferred Term will be counted only once within the SOC and PT

Coding dictionnary: MedDRA version xx.x (Month year)

Data source(s): addmain.xxxx (Date time)

Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)

Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name

#### This mock table is used for the following tables:

Table 14.3.3.2: Any Unsolicited TEAE during Period 1 by SOC, PT and Relatedness - SAF Analysis Set
Table 14.3.3.3: Any Unsolicited TEAE during Period 1 and Period 2 by SOC, PT and Relatedness - SAF Analysis Set
Table 14.3.3.4: Any Unsolicited TEAE during Period 2 by SOC, PT and Relatedness - SAF Analysis Set
Table 14.3.3.5: Any Unsolicited TEAE during Period 2 and Period 3 by SOC, PT and Relatedness - SAF Analysis Set
Table 14.3.3.6: Any Unsolicited TEAE during Period 3 by SOC, PT and Relatedness - SAF Analysis Set
Table 14.3.3.7: Any Unsolicited TEAE during Period 3 and Period 4 by SOC, PT and Relatedness - SAF Analysis Set
Table 14.3.4.1: Any Solicited AE by SOC/PT and Maximum Severity during Period 1 - SAF Analysis Set
Table 14.3.4.2: Any Unsolicited TEAE by SOC/PT and Maximum Severity during Period 1 - SAF Analysis Set
Table 14.3.4.3: Any Unsolicited TEAE by SOC/PT and Maximum Severity during Period 1 - SAF Analysis Set
Table 14.3.4.4: Any Unsolicited TEAE by SOC/PT and Maximum Severity during Period 1 and Period 2 - SAF Analysis Set
Table 14.3.4.5: Any Unsolicited TEAE by SOC/PT and Maximum Severity during Period 2 - SAF Analysis Set
Table 14.3.4.6: Any Unsolicited TEAE by SOC/PT and Maximum Severity during Period 2 and Period 3 - SAF Analysis Set
Table 14.3.4.7: Any Unsolicited TEAE by SOC/PT and Maximum Severity during Period 3 - SAF Analysis Set
Table 14.3.4.8: Any Unsolicited TEAE by SOC/PT and Maximum Severity during Period 3 - SAF Analysis Set
Table 14.3.8: Any Unsolicited TEAE by SOC/PT and Maximum Severity during Period 3 - SAF Analysis Set
Table 14.3.8: Any Unsolicited TEAE by SOC/PT and Maximum Severity during Period 3 and Period 4 - SAF Analysis Set
Table 14.3.8: Any SAE by SOC, PT and Relatedness across all Periods - SAF Analysis Set




| Document Number | or Drainet | Idontification | CIDADA | CDT CCD 001 |
|-----------------|------------|-----------------|--------|-------------|
| Document Number | or Project | identification. | CIDARA | CD1-C25-001 |


# **Mock Tables and Figures**

# List of Figures

| n° | Efficacy Results | IA |
|---|---|---|
| 14.2.1.1.1 | Primary efficacy analysis – Box Plots for VL-AUC from qRT-PCR – PP Analysis Set | Х |
| 14.2.1.1.2 | Primary efficacy analysis – Plots of Mean VL-AUC from qRT-PCR over time – PP Analysis Set | Х |
| 14.2.1.2.1.1 | Primary efficacy analysis – Box Plots for VL-AUC from qRT-PCR – ITT Analysis Set | |
| 14.2.1.2.1.2 | Primary efficacy analysis – Plots of Mean VL-AUC from qRT-PCR over time – ITT Analysis Set | |
| 14.2.1.2.2.1 | Primary efficacy analysis – Box Plots for VL-AUC from qRT-PCR – ITT-I Analysis Set | |
| 14.2.1.2.2.2 | Primary efficacy analysis – Plots of Mean VL from qRT-PCR over time – ITT-I Analysis Set | |
| 14.2.2.1 | Box Plots for Peak Viral Load from qRT-PCR – PP Analysis Set | Х |
| 14.2.2.2 | Box Plots for Peak Viral Load from qRT-PCR – ITT-I Analysis Set | |
| 14.2.3.1 | Time to Confirmed Negative Test by qRT-PCR – PP Analysis Set | |
| 14.2.3.2 | Time to Confirmed Negative Test by qRT-PCR – ITT-I Analysis Set | |
| 14.2.4.1.1 | Box Plots for VL-AUC from Viral Culture – PP Analysis Set | |
| 14.2.4.1.2 | Plots of Mean VL from Viral Culture over time – PP Analysis Set | |
| 14.2.4.2.1 | Box Plots for VL-AUC from Viral Culture – ITT-I Analysis Set | |
| 14.2.4.2.2 | Plots of Mean VL from Viral Culture over time – ITT-I Analysis Set | |
| 14.2.5.1 | Box Plots for Peak Viral Load from Viral Culture – PP Analysis Set | |
| 14.2.5.2 | Box Plots for Peak Viral Load from Viral Culture – ITT-I Analysis Set | |
| 14.2.6.1 | Time to Confirmed Negative Test by from Viral Culture – PP Analysis Set | Х |
| 14.2.6.2 | Time to Confirmed Negative Test by from Viral Culture – ITT-I Analysis Set | |
| 14.2.7.1.1 | Box Plots for TSS-AUC- PP Analysis Set | Х |
| 14.2.7.1.2 | Plots of Mean TSS over time – PP Analysis Set | Х |
| 14.2.7.2.1 | Box Plots for TSS-AUC – ITT-I Analysis Set | |



| <b>Document Number or Pro</b> | ject Identification: | CIDARA | CDT-CSP-001 |
|---|---|---|---|
|---|---|---|---|

# **Mock Tables and Figures**

| 14.2.7.2.2 | Plots of Mean TSS over time – ITT-I Analysis Set | |
|---|---|---|
| 14.2.8.1 | Box Plots for Peak Total Clinical Symptoms Score – PP Analysis Set | Х |
| 14.2.8.2 | Box Plots for Peak Total Clinical Symptoms Score – ITT-I Analysis Set | |
| 14.2.9.1 | Plots of Mean Peak Daily Total Clinical Symptoms Score over time – PP Analysis Set | |
| 14.2.9.2 | Plots of Mean Peak Daily Total Clinical Symptoms Score over time – ITT-I Analysis Set | |
| 14.2.10.1 | Time to Symptom Resolution – PP Analysis Set | Х |
| 14.2.10.2 | Time to Symptom Resolution – ITT-I Analysis Set | |
| 14.3.1 | Laboratory Safety: Plots of Mean Raw Values over time – SAF Analysis Set | |




# **Mock Tables and Figures**

Figure 14.2.1.1.1: Primary efficacy analysis - Box Plots for VL-AUC from qRT-PCR

PP Analysis Set



Data source(s): addmain.xxxx (Date time)
Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)
Program: /Study/tlf/tf/pgm/pgm\_name.sas Date time / run Date time by Stat\_name





## **Mock Tables and Figures**

### This mock figure is used for the following figures:

```
Figure 14.2.1.2.1.1: Primary efficacy analysis - Box Plots for VL-AUC from qRT-PCR - ITT Analysis Set
Figure 14.2.1.2.2.1: Primary efficacy analysis - Box Plots for VL-AUC from qRT-PCR - ITT-I Analysis Set
Figure 14.2.2.1: Box Plots for Peak Viral Load from qRT-PCR - PP Analysis Set
Figure 14.2.2.2: Box Plots for Peak Viral Load from qRT-PCR - ITT-I Analysis Set
Figure 14.2.4.1.1: Box Plots for VL-AUC from Viral Culture - PP Analysis Set
Figure 14.2.4.2.1: Box Plots for VL-AUC from Viral Culture - ITT-I Analysis Set
Figure 14.2.5.1: Box Plots for Peak Viral Load from Viral Culture - PP Analysis Set
Figure 14.2.5.2: Box Plots for Peak Viral Load from Viral Culture - ITT-I Analysis Set
Figure 14.2.7.1.1: Box Plots for TSS-AUC - PP Analysis Set
Figure 14.2.7.2.1: Box Plots for TSS-AUC - ITT-I Analysis Set
Figure 14.2.8.1: Box Plots for Peak Total Clinical Symptoms Score - PP Analysis Set
Figure 14.2.8.2: Box Plots for Peak Total Clinical Symptoms Score - ITT-I Analysis Set
```


# **Mock Tables and Figures**

Figure 14.2.1.1.2: Primary efficacy analysis - Plots of Mean VL-AUC from RT-qPCR over time

PP Analysis Set



Data source(s): addmain.xxxx (Date time)
Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)
Program: /Study/tlf/tf/pgm/pgm\_name.sas Date time / run Date time by Stat\_name




## **Mock Tables and Figures**

### This mock figure is used for the following figures:

```
Figure 14.2.1.2.1.2: Primary efficacy analysis - Plots of Mean VL-AUC from RT-qPCR over time - ITT Analysis Set
Figure 14.2.1.2.2.2: Primary efficacy analysis - Plots of Mean VL-AUC from RT-qPCR over time - ITT-I Analysis Set
Figure 14.2.4.1.3: Plots of Mean VL from Viral Culture over time - PP Analysis Set
Figure 14.2.4.2.2: Plots of Mean VL from Viral Culture over time - ITT-I Analysis Set
Figure 14.2.7.1.3: Plots of Mean TSS over time - PP Analysis Set
Figure 14.2.7.2.2: Plots of Mean TSS over time - ITT-I Analysis Set
Figure 14.2.9.1: Plots of Mean Peak Daily Total Clinical Symptoms Score over time - PP Analysis Set
Figure 14.2.9.2: Plots of Mean Peak Daily Total Clinical Symptoms Score over time - ITT-I Analysis Set
Figure 14.3.1: Laboratory Safety: Plots of Mean Raw Values over time - SAF Analysis Set
```




# **Mock Tables and Figures**

Figure 14.2.3.1: Time to Confirmed Negative Test by qRT-PCR - PP Analysis Set

PP Analysis Set



Data source(s): addmain.xxxx (Date time)
Analysis dataset(s): adsmain.adxxx (Date time) adsmain.adxxx (Date time)
Program: /Study/tlf/tf/pgm/pgm name.sas Date time / run Date time by Stat name




| <b>Document Number or Pro</b> | ect Identification: | CIDARA | CDT-CSP-003 |
|-------------------------------|---------------------|--------|-------------|

# **Mock Tables and Figures**

## This mock figure is used for the following figures:

Figure 14.2.3.2: Time to Confirmed Negative Test by qRT-PCR - ITT-I Analysis Set

Figure 14.2.6.1: Time to Confirmed Negative Test by from Viral Culture - PP Analysis Set

Figure 14.2.6.2: Time to Confirmed Negative Test by from Viral Culture - ITT-I Analysis Set

Figure 14.2.10.1: Time to Symptom Resolution - PP Analysis Set

Figure 14.2.10.2: Time to Symptom Resolution - ITT-I Analysis Set


# **DocuSign**

## **Certificate Of Completion**

Envelope Id: B29BDF7A296345A5AD00D75C78B3CEAE

Subject: CIDARA\_CDT-CSP-001\_SAP V2 and Mock Tables V1\_Final\_25Jul23

Source Envelope:

Document Pages: 107 Certificate Pages: 3

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-08:00) Pacific Time (US & Canada)

Status: Completed

Envelope Originator: Joaquin Sosa

6310 Nancy Ridge Dr

STE 101

San Diego, CA 92121 jsosa@cidara.com

IP Address: 136.49.202.34

Sent: 7/25/2023 8:01:44 AM

Viewed: 7/25/2023 8:11:39 AM

Signed: 7/25/2023 8:12:28 AM

### **Record Tracking**

Status: Original

7/25/2023 7:57:06 AM

Holder: Joaquin Sosa jsosa@cidara.com

Location: DocuSign

**Timestamp** 

### **Signer Events**

Antoinette Anger

antoinette.anger@vennlife.com

Security Level: Email, Account Authentication

(Required)

### Signature

D

Signatures: 3

Initials: 0

-DocuSigned by:

Antoinette Anger

Signer Name: Antoinette Anger Signing Reason: I am the author of this document Signing Time: 25-Jul-2023 | 8:12:21 AM PDT

—D8AB006C654B4E9CB5F4CE85D0841495

Signature Adoption: Pre-selected Style

Signature ID:

D8AB006C-654B-4E9C-B5F4-CE85D0841495

Using IP Address: 78.194.28.65

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

## **Electronic Record and Signature Disclosure:**

Accepted: 7/25/2023 8:11:39 AM

ID: 5e08b13b-1649-4407-a813-45926b79c576

Elodie Blondiaux

Elodie.Blondiaux@vennlife.com

Security Level: Email, Account Authentication

(Required)

Elodie Blandiaux

Sent: 7/25/2023 8:01:44 AM Viewed: 7/25/2023 8:12:49 AM

Signed: 7/25/2023 8:13:44 AM

Signature Adoption: Pre-selected Style

Signature ID:

4832F141-BED9-40A2-A126-AB01E747A040

Using IP Address: 88.167.158.14

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):
I have reviewed this document

### **Electronic Record and Signature Disclosure:**

Accepted: 7/25/2023 8:12:49 AM

ID: 447af0c8-cdf0-4053-8093-05bdeef5a247

**Signer Events** 

Ozlem Equils, MD oequils@cidara.com

Security Level: Email, Account Authentication

(Required)

**Signature** 

U

DocuSigned by:

Signer Name: Ozlem Equils, MD Signing Reason: I approve this document Signing Time: 25-Jul-2023 | 8:08:25 AM PDT

8C319F80E19A475B89044981B91CEB55

Signature Adoption: Drawn on Device

Signature ID:

8C319F80-E19A-475B-8904-4981B91CEB55

Using IP Address: 98.207.229.100

Signed using mobile

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 7/25/2023 8:07:43 AM

ID: b652a38c-e19d-455d-9b4e-3c470ff32027

| In Person Signer Events | Signature | Timestamp |
|------------------------------------|-----------|----------------------------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Hardeep Johal<br>h.johal@hvivo.com | COPIED | Sent: 7/25/2023 8:01:45 AM |

h.johal@hvivo.com Project Manager

**Witness Events** 

**Notary Events** 

**Envelope Sent** Certified Delivered Signing Complete

Completed

Security Level: Email, Account Authentication

(Required)

**Electronic Record and Signature Disclosure:** 

Accepted: 8/26/2022 2:21:35 AM

**Envelope Summary Events** 

ID: b236cd41-3d0a-41d5-8052-8ae9eae30d18

| Signature | Timestamp |
|-------------------------|----------------------|
| Signature | Timestamp |
| <b>0</b> / / | |
| Status | Timestamps |
| Status Hashed/Encrypted | 7/25/2023 8:01:45 AM |
| | • |

7/25/2023 8:13:44 AM

**Timestamp** 

Sent: 7/25/2023 8:01:45 AM

Viewed: 7/25/2023 8:07:43 AM

Signed: 7/25/2023 8:08:27 AM

#### **Payment Events Status Timestamps**

Security Checked

**Electronic Record and Signature Disclosure** 

### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

By accepting this notice, I am documenting that I understand and approve the following:

- 1. When I sign documents or data electronically, I am accountable and responsible for all items thus signed.
- 2. I am to be held responsible for all actions initiated under my electronic signature.
- 3. I will use my electronic signature only for those assigned tasks that I have the education, training, and experience to perform.

I will comply with the US FDA 21 CFR Part 11 and EU Annex 11 security rules for Cidara Therapeutics use of electronic signatures as follows:

- 1. I will not share passwords and/or identification codes used to log into a system or to manifest an electronic signature for Cidara Therapeutics documents.
- 2. I will immediately notify Cidara Therapeutics of any loss of misuse of passwords and/or identification codes which may have been used to log into a system or to manifest an electronic signature for Cidara Therapeutics documents.